# Protocol CMUH110-REC2-070

# The Effect of Lactobacillus Delbrueckii Subsp. Bulgaricus on Human's Weight Reduction

Document type: Study Protocol with Statistical Analysis Plan (SAP)

Version number 02

Document status: Final report

Release date 03-Feb-2023

Author:

Number of pages: 28

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 2/28 |

## **Table of contents**

| Table of contents | 2 |
|--------------------|----|
| Background | 3 |
| Methods and Design | 4 |
| Results | 7 |
| Appendix | 14 |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 3/28 |

### **Background**

In recent years, probiotic supplements have become increasingly popular in daily life for preventing diarrhea, easing vaginal and urinary infections, or preventing autoimmune diseases [1–3]. Probiotics cause the formation of a properly balanced gut bacterial population, with balance between pathogens and the bacteria necessary for normal functioning of the organism, and may improve immune system function and nutrient absorption. Recently, the gut microbiota was found to be involved in various metabolic pathways and energy balance regulation [4, 5]. The composition of the gut microbiota differs between obese and normal weight individuals [6, 7]. Dietary alteration of the gut microbiome is a target for treating obesity [8]. However, clinical trials examining the influence of probiotics on obesityrelated factors have yielded inconsistent outcomes. Some studies have demonstrated weight loss in participants supplemented with lactobacilli and bifidobacteria, even while maintaining their normal diet and lifestyle over the study's duration [9,10]. In a 12-week trial, participants consuming L. gasseri experienced significant reductions in visceral fat, body mass index, waist and hip circumference, and body fat mass compared to the control group [11]. Conversely, another trial involving *L. rhamnosus* supplementation alongside an energy-restricted diet did not significantly impact weight loss in all participants but showed a reduction in weight in females [12]. Systematic review, encompassing 19 randomized trials with 1,412 participants, revealed diverse outcomes [13]. Some studies report significant decreases in body weight and/or body fat with probiotics, while others indicate no effect or even increased body weight. It suggests that specific probiotics have the potential to serve as health supplements for treating or preventing obesity and overweight.

Lactobacillus is a type of lactic acid bacterium commonly found in the human gastrointestinal tract and in fermented dairy products such as cheese, yogurt, and kefir [14]. The isolation of specific probiotic strains for targeted application is a strategy for improving the efficacy of probiotic supplements. Some species of Lactobacillus, such as L. gasseri and L. rhamnosus, have been evaluated for inducing weight loss [15]. Lactobacillus delbrueckii ssp. bulgaricus (L. bulgaricus) is one of the most common lactobacilli starters used in the manufacture of a large variety of fermented milk products. L. bulgaricus is reported to exhibit an outstanding inhibitory effect on pancreatic lipase activity in vitro and effectively managed the fat and weight accumulation and reversed the increased blood lipid, sugar, and insulin levels caused by a high-fat diet in mice [16]. Our hypothesis posits that L. bulgaricus can contribute to the reduction of body weight and alleviate health risk factors associated with obesity in overweight individuals. Thus, the objective of this study was to examine the effectiveness of daily L. bulgaricus supplementation in weight management among overweight participants. The primary goal is to evaluate its impact on lowering body weight and addressing health risk factors related to obesity, including blood lipid levels, sugar regulation, and insulin levels.

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 4/28 |

## **Methods and Design**

#### **Participants:**

The participants were recruited from the patients of Endocrinology and Metabolism Department at China Medical University Hospital, followed by the verification of inclusion and exclusion criteria through interviews. The inclusion criteria comprised: (1) age  $\geq 20$ years old; (2) overweight (BMI  $\geq$  23) or body fat percentage  $\geq$  25% for males and  $\geq$  30% for females; (3) having any of the following risk factors: atherosclerotic cardiovascular disease (ASCVD), type 2 diabetes, age  $\geq$  45 years for males,  $\geq$  55 years for females or postmenopausal, hypertension, dyslipidemia (total cholesterol(CHOL) > 200 mg/dL or low-density lipoprotein cholesterol (LDL-C) > 130 mg/dL or triglycerides (TG) > 130 mg/dL), highdensity lipoprotein cholesterol (HDL-C) < 40 mg/dL; (4) if routinely taking medication for lowering blood glucose, blood pressure, or lipid levels, there should not be significant dosage changes within the past three months; (5) being willing to participate after receiving an explanation from the physician, completing the trial plan, and signing the consent form. The exclusion criteria included: (1) history of diabetic ketoacidosis; (2) medical records indicating the occurrence of cerebrovascular disease, acute myocardial infarction, coronary artery bypass surgery, placement of coronary artery stents, or peripheral vascular disease within the last 6 months; (3) occurrence of acute infectious diseases within the last month and antibiotic use for > 7 days; (4) short-term use of steroids, NSAIDs, immunosuppressive drugs, interferons, immunomodulators, or any changes in the dose of long-term medications within the last month; (5) use of any weight-loss drugs in the last three months (including Orlistat, Lorcaserin, liraglutide); (6) history of any cancer or undergoing cancer treatment in the past 5 years; (7) abnormal liver function (GOT or GPT greater than 3 times the normal upper limit) or liver cirrhosis; (8) impaired kidney function (eGFR < 30 mL/min/1.73 m<sup>2</sup>); (9) history of alcohol abuse; (10) participation in any other interventional clinical research within the last month; (11) pregnant and breastfeeding women; (12) history of allergy to the investigational product; (13) participants deemed unsuitable for inclusion by the principal investigator.

### **Study Design and Intervention:**

Enrolled participants were randomly divided into probiotics group or placebo group. Seventeen and 19 participants were respectively assigned to the placebo group and the probiotics group. The probiotics we used were in the form of 100mg L. bulgaricus powder packets, each containing 1x10^8 CFU of probiotics (TCI CO., Taipei, Taiwan). Initially (day 1), participants underwent measurements for weight, body fat, and BMI, and fasting blood

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 5/28 |

samples were collected. Subsequently, each participant received one package of either probiotic or a placebo sample, along with drinking water on the same day. From that point onward, participants self-administered one package of the sample daily for 12 weeks and the participants' sample consumption and physical conditions were tracked by the research assistants weekly. Throughout the study duration, participants maintained their regular diet and lifestyle. At the endpoint (day 84), weight, body fat, and BMI were measured, and fasting blood samples were collected again. Weight and body fat were measured with Karada Scan 216 (OMRON, Kyoto, Japan). Alanine aminotransferase (ALT), aspartate aminotransferase (AST), blood urea nitrogen (BUN), creatinine (CRE), CHOL, HDL-C, LDL-C, TG, hemoglobin A1c (HbA1c), and Glucose-Ante Cibum (Glu-AC) levels were analyzed and reported by Laboratory Medicine in Chinese Medical University Hospital (Taichung, Taiwan). Data were expressed as the mean ± standard error of the mean (SEM). Statistical significance between groups were done by student paired t-test or Mann-Whitney test. P-values lower than 0.05 were considered statistically significant.

#### **Data Analysis:**

The statistical analysis was conducted using GraphPad's unpaired independent samples t-test, with significance set at \*P<0.05.

#### Flow Diagram of the study:



| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 6/28 |

| Group | Placebo | | Probiotics | |
|---------------------|---------|-------|------------|--------|
| | Mean | SD | Mean | SD |
| Age, years | 41.38 | 12.71 | 41.56 | 10.92 |
| Gender, male/female | 7/6 | | 12/6 | |
| Weight, kg | 78.69 | 15.64 | 80.77 | 15.11 |
| Body fat, % | 32.08 | 6.65 | 30.84 | 5.26 |
| BMI | 29.32 | 5.40 | 28.89 | 3.59 |
| ALT, U/L | 26.00 | 15.37 | 32.63 | 18.96 |
| AST, U/L | 21.45 | 10.62 | 23.36 | 7.44 |
| BUN, mg/dL | 13.10 | 2.69 | 13.67 | 2.94 |
| CRE, mg/dL | 0.80 | 0.14 | 0.83 | 0.15 |
| CHOL, mg/dL | 182.18 | 43.04 | 201.60 | 40.97 |
| HDL-C, mg/dL | 46.82 | 5.82 | 48.50 | 16.26 |
| LDL-C, mg/dL | 122.82 | 42.15 | 111.01 | 30.40 |
| TG, mg/dL | 139.62 | 52.18 | 220.94 | 173.92 |
| HbA1c, % | 5.80 | 0.83 | 6.17 | 1.07 |
| Glu-AC, mg/dL | 93.45 | 16.92 | 109.06 | 34.13 |

Table 1: Analysis of Baseline Values of the Participants

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 7/28 |

## **Results**



Figure 1: Changes in Body Composition

Placebo represents the placebo control group, and Probiotics represents the probiotics experimental group. The changes in body weight (A), body fat (B), and BMI (C) before and after consumption were calculated and expressed as a percentage of the initial values. No significant differences were observed between the two groups.



Figure 2: Changes in Blood Sugar Indices

Placebo represents the placebo control group, and Probiotics represents the probiotics experimental group. The changes in fasting blood glucose (GLU-AC) before and after sample consumption (A) and changes in glycated hemoglobin (HbA1c) expressed as a percentage of the initial values (B) were calculated. No significant differences were observed

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 8/28 |

between the two groups.



Figure 3: Changes in Blood Lipids

Placebo represents the placebo control group, and Probiotics represents the probiotics experimental group. The changes in total cholesterol (CHOL) (A), triglycerides (TG) (B), high-density lipoprotein cholesterol (HDL) (C), and low-density lipoprotein cholesterol (LDL-C) (D) before and after sample consumption were calculated. No significant differences were observed between the two groups. In the probiotics group, 65% of participants showed a decrease in TG concentration, while the placebo group had a decrease rate of 18%.

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 9/28 |



Figure 4: Changes in Liver and Kidney Function

Placebo represents the placebo control group, and Probiotics represents the probiotics experimental group. The changes in liver function indicators, aspartate aminotransferase (AST) (A) and alanine aminotransferase (ALT) (B), as well as kidney function indicators, creatinine (CRE) (C) and blood urea nitrogen (BUN) (D), before and after sample consumption were calculated. No significant differences were observed between the two groups.

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 10/28 |

Table 2: Comparative Analysis of Blood Biochemical Indices Before and After the Experiment and Changes Before and After

| Variables | | Probiotics | Placebo | |
|---|---|---|---|---|
| | | Mean ± SEM | Mean ± SEM | P-valueb |
| ALT (U/L) | Pre | $32.00 \pm 4.495$ | $31.00 \pm 6.454$ | 0.9897 |
| | Post | $28.12 \pm 4.853$ | $37.69 \pm 7.946$ | 0.7713 |
| | Change | $-3.882 \pm 3.461$ | $6.692 \pm 6.747$ | 0.5075 |
| | P-valuea | 0.2462 | 0.3799 | |
| AST (U/L) | Pre | 24.31 ± 1.886 | 22.38 ± 3.054 | 0.3909 |
| | Post | $22.44 \pm 2.238$ | $25.85 \pm 4.366$ | 0.9053 |
| | Change | $-1.875 \pm 1.530$ | $3.462 \pm 2.043$ | 0.34 |
| | P-valuea | 0.0708 | 0.1367 | |
| BUN (mg/dL) | Pre | $13.82 \pm 0.6765$ | 13.17 ± 0.8242 | 0.9267 |
| | Post | $12.88 \pm 0.8985$ | $12.67 \pm 0.7914$ | 0.9694 |
| | Change | $-0.6250 \pm 0.7465$ | $-0.5000 \pm 0.8118$ | >0.999 |
| | P-valuea | 0.5256 | 0.6504 | |
| CRE (mg/dL) | Pre | $0.8241 \pm 0.03584$ | $0.7962 \pm 0.0443$ | 0.907 |
| | Post | $0.8775 \pm 0.04979$ | $0.7915 \pm 0.04273$ | 0.6543 |
| | Change | $0.0475 \pm 0.02713$ | $-0.004615 \pm 0.02087$ | 0.34 |
| | P-valuea | 0.0535 | 0.8262 | |
| CHOL (mg/dL) | Pre | $200.7 \pm 10.33$ | $186.9 \pm 11.49$ | 0.67 |
| | Post | $204.6 \pm 12.42$ | $186.3 \pm 10.20$ | 0.0719 |
| | Change | $3.882 \pm 7.086$ | $-0.6154 \pm 3.852$ | 0.5075 |
| | P-valuea | 0.6526 | 0.8535 | |
| Glu-AC (mg/dL) | Pre | $109.3 \pm 7.834$ | $91.77 \pm 4.590$ | 0.3871 |
| | Post | $100.7 \pm 9.383$ | $91.69 \pm 6.466$ | 0.5854 |
| | Change | $1.389 \pm 2.332$ | $-0.07692 \pm 2.962$ | 0.7803 |
| | P-valuea | 0.6183 | 0.6846 | |
| HbA1c (%) | Pre | $6.124 \pm 0.2559$ | $5.800 \pm 0.2295$ | 0.8619 |
| | Post | $6.407 \pm 0.3149$ | $5.931 \pm 0.3175$ | 0.6367 |
| | Change | $0.2067 \pm 0.05893$ | $0.1308 \pm 0.09765$ | 0.4821 |
| | P-valuea | 0.0029 | 0.2061 | |
| HDL-C (mg/dL) | Pre | $48.55 \pm 3.820$ | $46.82 \pm 1.613$ | 0.3643 |
| | Post | $47.38 \pm 3.125$ | $46.43 \pm 1.798$ | 0.4656 |
| | Change | $-0.0125 \pm 1.362$ | $-0.3923 \pm 1.590$ | 0.9872 |
| | P-valuea | 0.4037 | 0.7227 | |
| LDL-C (mg/dL) | Pre | 113.0 ± 7.399 | 122.8 ± 12.17 | 0.4531 |
| | Post | $119.0 \pm 5.992$ | $112.4 \pm 8.306$ | 0.5874 |

| | | | IRB/REC No.: | CMUH110-REC2<br>-070 |
|---|---|---|---|---|
| | | | Page No.: | 11/28 |
| | Change | 6.012 ± 4.366 | $-12.04 \pm 6.323$ | 0.0946 |
| | P-valuea | 0.4586 | 0.0923 | |
| TG (mg/dL) | Pre | $220.9 \pm 42.18$ | $139.6 \pm 14.47$ | 0.5469 |
| | Post | $199.9 \pm 40.46$ | $177.4 \pm 36.55$ | 0.907 |
| | Change | $-21.00 \pm 11.61$ | $37.77 \pm 34.12$ | 0.0555 |
| | P-valuea | 0.1075 | 0.1577 | |

P-valuea paired t-test (Pre and Post groups)

P-valueb unpaired t-test (Probiotics and Placebo groups)

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 12/28 |



Figure 5: Changes in Lipids Carried by Serum Lipoproteins

Placebo represents the placebo control group, and Probiotics represents the probiotics experimental group. Individual comparisons of changes in lipids carried by serum lipoproteins before and after sample consumption are depicted. The size of the points in the scatter plot (-log10 p values) and the color (log2 fold change denoted as log2FC, with red indicating positive correlation changes and blue indicating negative correlation changes) are used to distinguish between inter-group differences and trends. Serum very low-density lipoprotein (VLDL), low-density lipoprotein (LDL), and high-density lipoprotein (HDL) have the ability to carry cholesterol (Chol), lipids, cholesterol esters (CE), and triglycerides (TG) individually. The experimental data indicate that probiotics upregulate the content of

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 13/28 |

lipids carried by HDL (Chol:Lipid and CE:Lipid). Simultaneously, there is a significant decrease in the total amount of lipids carried by VLDL (L-VLDL, XL-VLDL, XXL-VLDL). Additionally, there is a significant decrease in triglycerides (TG) carried by both VLDL and HDL.

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 14/28 |

# **Appendix**

Figure 5: Extracted Meaningful Components from Metabolomic Analysis Results, Other Results Provided in the Appendix  $^\circ$ 

Table 3: List of Name Abbreviations and Units

| Excel column name | Biomarker name | Unit |
|---|---|---|
| Total-C | Total cholesterol | mmol/l |
| non-HDL-C | Total cholesterol minus HDL-C | mmol/l |
| Remnant-C | Remnant cholesterol (non-HDL, non-LDL -cholesterol) | mmol/l |
| VLDL-C | VLDL cholesterol | mmol/l |
| Clinical LDL-C | Clinical LDL cholesterol | mmol/l |
| LDL-C | LDL cholesterol | mmol/l |
| HDL-C | HDL cholesterol | mmol/l |
| Total-TG | Total triglycerides | mmol/l |
| VLDL-TG | Triglycerides in VLDL | mmol/l |
| LDL-TG | Triglycerides in LDL | mmol/l |
| HDL-TG | Triglycerides in HDL | mmol/l |
| Total-PL | Total phospholipids in lipoprotein particles | mmol/l |
| VLDL-PL | Phospholipids in VLDL | mmol/l |
| LDL-PL | Phospholipids in LDL | mmol/l |
| HDL-PL | Phospholipids in HDL | mmol/l |
| Total-CE | Total esterified cholesterol | mmol/l |
| VLDL-CE | Cholesteryl esters in VLDL | mmol/l |
| LDL-CE | Cholesteryl esters in LDL | mmol/l |
| HDL-CE | Cholesteryl esters in HDL | mmol/l |
| Total-FC | Total free cholesterol | mmol/l |
| VLDL-FC | Free cholesterol in VLDL | mmol/l |
| LDL-FC | Free cholesterol in LDL | mmol/l |
| HDL-FC | Free cholesterol in HDL | mmol/l |
| Total-L | Total lipids in lipoprotein particles | mmol/l |
| VLDL-L | Total lipids in VLDL | mmol/l |
| LDL-L | Total lipids in LDL | mmol/l |
| HDL-L | Total lipids in HDL | mmol/l |
| Total-P | Total concentration of lipoprotein particles | mmol/l |
| VLDL-P | Concentration of VLDL particles | mmol/l |
| LDL-P | Concentration of LDL particles | mmol/l |
| HDL-P | Concentration of HDL particles | mmol/l |
| VLDL size | Average diameter for VLDL particles | nm |
| LDL size | Average diameter for LDL particles | nm |
| HDL size | Average diameter for HDL particles | nm |
| Phosphoglyc | Phosphoglycerides | mmol/l |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 15/28 |

| TG/PG | Ratio of triglycerides to phosphoglycerides | ratio |
|---|---|---|
| Cholines | Total cholines | mmol/l |
| Phosphatidylc | Phosphatidylcholines | mmol/l |
| Sphingomyelins | Sphingomyelins | mmol/l |
| ApoB | Apolipoprotein B | g/l |
| ApoA1 | Apolipoprotein Al | g/l |
| ApoB/ApoA1 | Ratio of apolipoprotein B to apolipoprotein A1 | ratio |
| Total-FA | Total fatty acids | mmol/l |
| Unsaturation | Degree of unsaturation | degree |
| Omega-3 | Omega-3 fatty acids | mmol/l |
| Omega-6 | Omega-6 fatty acids | mmol/l |
| PUFA | Polyunsaturated fatty acids | mmol/l |
| MUFA | Monounsaturated fatty acids | mmol/l |
| SFA | Saturated fatty acids | mmol/l |
| LA | Linoleic acid | mmol/l |
| DHA | Docosahexaenoic acid | mmol/l |
| Omega-3 % | Ratio of omega-3 fatty acids to total fatty acids | % |
| Omega-6 % | Ratio of omega-6 fatty acids to total fatty acids | % |
| PUFA % | Ratio of polyunsaturated fatty acids to total fatty acids | % |
| MUFA % | Ratio of monounsaturated fatty acids to total fatty acids | % |
| SFA % | Ratio of saturated fatty acids to total fatty acids | % |
| LA % | Ratio of linoleic acid to total fatty acids | % |
| DHA % | Ratio of docosahexaenoic acid to total fatty acids | % |
| PUFA/MUFA | Ratio of polyunsaturated fatty acids to monounsaturated fatty acids | ratio |
| Omega-6/Omega-3 | Ratio of omega-6 fatty acids to omega-3 fatty acids | ratio |
| Ala | Alanine | mmol/l |
| Gln | Glutamine | mmol/l |
| Gly | Glycine | mmol/l |
| His | Histidine | mmol/l |
| Total BCAA | Total concentration of branched-chain amino acids (leucine + isoleucine + valine) | mmol/l |
| Ile | Isoleucine | mmol/l |
| Leu | Leucine | mmol/l |
| Val | Valine | mmol/l |
| Phe | Phenylalanine | mmol/l |
| Tyr | Tyrosine | mmol/l |
| Glucose | Glucose | mmol/l |
| Lactate | Lactate | mmol/l |
| Pyruvate | Pyruvate | mmol/l |
| Citrate | Citrate | mmol/l |
| Glycerol | Glycerol | mmol/l |
| bOHbutyrate | 3-Hydroxybutyrate | mmol/l |
| Acetate | Acetate | mmol/l |
| Acetoacetate | Acetoacetate | mmol/l |
| Acetone | Acetone | mmol/l |
| Creatinine | Creatinine | $\mu$ mol/l |
| > | 1 | 1 |

| IRB/REC No.: | CMUH110-REC2 |
|--------------|--------------|
| | -070 |
| Page No.: | 16/28 |

| Albumin | Albumin | g/l |
|---|---|---|
| GlycA | Glycoprotein acetyls | mmol/l |
| XXL-VLDL-P | Concentration of chylomicrons and extremely large VLDL particles | mmol/l |
| XXL-VLDL-L | Total lipids in chylomicrons and extremely large VLDL | mmol/l |
| XXL-VLDL-PL | Phospholipids in chylomicrons and extremely large VLDL | mmol/l |
| XXL-VLDL-C | Cholesterol in chylomicrons and extremely large VLDL | mmol/l |
| XXL-VLDL-CE | Cholesteryl esters in chylomicrons and extremely large VLDL | mmol/l |
| XXL-VLDL-FC | Free cholesterol in chylomicrons and extremely large VLDL | mmol/l |
| XXL-VLDL-TG | Triglycerides in chylomicrons and extremely large VLDL | mmol/l |
| XL-VLDL-P | Concentration of very large VLDL particles | mmol/l |
| XL-VLDL-L | Total lipids in very large VLDL | mmol/l |
| XL-VLDL-PL | Phospholipids in very large VLDL | mmol/l |
| XL-VLDL-C | Cholesterol in very large VLDL | mmol/l |
| XL-VLDL-CE | Cholesteryl esters in very large VLDL | mmol/l |
| XL-VLDL-FC | Free cholesterol in very large VLDL | mmol/l |
| XL-VLDL-TG | Triglycerides in very large VLDL | mmol/l |
| L-VLDL-P | Concentration of large VLDL particles | mmol/l |
| L-VLDL-L | Total lipids in large VLDL | mmol/l |
| L-VLDL-PL | Phospholipids in large VLDL | mmol/l |
| L-VLDL-C | Cholesterol in large VLDL | mmol/l |
| L-VLDL-CE | Cholesteryl esters in large VLDL | mmol/l |
| L-VLDL-FC | Free cholesterol in large VLDL | mmol/l |
| L-VLDL-TG | Triglycerides in large VLDL | mmol/l |
| M-VLDL-P | Concentration of medium VLDL particles | mmol/l |
| M-VLDL-L | Total lipids in medium VLDL | mmol/l |
| M-VLDL-PL | Phospholipids in medium VLDL | mmol/l |
| M-VLDL-C | Cholesterol in medium VLDL | mmol/l |
| M-VLDL-CE | Cholesteryl esters in medium VLDL | mmol/l |
| M-VLDL-FC | Free cholesterol in medium VLDL | mmol/l |
| M-VLDL-TG | Triglycerides in medium VLDL | mmol/l |
| S-VLDL-P | Concentration of small VLDL particles | mmol/l |
| S-VLDL-L | Total lipids in small VLDL | mmol/l |
| S-VLDL-PL | Phospholipids in small VLDL | mmol/l |
| S-VLDL-C | Cholesterol in small VLDL | mmol/l |
| S-VLDL-CE | Cholesteryl esters in small VLDL | mmol/l |
| S-VLDL-FC | Free cholesterol in small VLDL | mmol/l |
| S-VLDL-TG | Triglycerides in small VLDL | mmol/l |
| XS-VLDL-P | Concentration of very small VLDL particles | mmol/l |
| XS-VLDL-L | Total lipids in very small VLDL | mmol/l |
| XS-VLDL-PL | Phospholipids in very small VLDL | mmol/l |
| XS-VLDL-C | Cholesterol in very small VLDL | mmol/l |
| XS-VLDL-CE | Cholesteryl esters in very small VLDL | mmol/l |
| XS-VLDL-FC | Free cholesterol in very small VLDL | mmol/l |
| XS-VLDL-TG | Triglycerides in very small VLDL | mmol/l |
| IDL-P | Concentration of IDL particles | mmol/l |
| IDL-L | Total lipids in IDL | mmol/l |
| IDL-PL | Phospholipids in IDL | mmol/l |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 17/28 |

| IDL-C | Cholesterol in IDL | mmol/l |
|------------------|-------------------------------------------|--------|
| IDL-CE | Cholesteryl esters in IDL | mmol/l |
| IDL-CE<br>IDL-FC | Free cholesterol in IDL | |
| | | mmol/l |
| IDL-TG | Triglycerides in IDL | mmol/l |
| L-LDL-P | Concentration of large LDL particles | mmol/l |
| L-LDL-L | Total lipids in large LDL | mmol/l |
| L-LDL-PL | Phospholipids in large LDL | mmol/l |
| L-LDL-C | Cholesterol in large LDL | mmol/l |
| L-LDL-CE | Cholesteryl esters in large LDL | mmol/l |
| L-LDL-FC | Free cholesterol in large LDL | mmol/l |
| L-LDL-TG | Triglycerides in large LDL | mmol/l |
| M-LDL-P | Concentration of medium LDL particles | mmol/l |
| M-LDL-L | Total lipids in medium LDL | mmol/l |
| M-LDL-PL | Phospholipids in medium LDL | mmol/l |
| M-LDL-C | Cholesterol in medium LDL | mmol/l |
| M-LDL-CE | Cholesteryl esters in medium LDL | mmol/l |
| M-LDL-FC | Free cholesterol in medium LDL | mmol/l |
| M-LDL-TG | Triglycerides in medium LDL | mmol/l |
| S-LDL-P | Concentration of small LDL particles | mmol/l |
| S-LDL-L | Total lipids in small LDL | mmol/l |
| S-LDL-PL | Phospholipids in small LDL | mmol/l |
| S-LDL-C | Cholesterol in small LDL | mmol/l |
| S-LDL-CE | Cholesteryl esters in small LDL | mmol/l |
| S-LDL-FC | Free cholesterol in small LDL | mmol/l |
| S-LDL-TG | Triglycerides in small LDL | mmol/l |
| XL-HDL-P | Concentration of very large HDL particles | mmol/l |
| XL-HDL-L | Total lipids in very large HDL | mmol/l |
| XL-HDL-PL | Phospholipids in very large HDL | mmol/l |
| XL-HDL-C | Cholesterol in very large HDL | mmol/l |
| XL-HDL-CE | Cholesteryl esters in very large HDL | mmol/l |
| XL-HDL-FC | Free cholesterol in very large HDL | mmol/l |
| XL-HDL-TG | Triglycerides in very large HDL | mmol/l |
| L-HDL-P | Concentration of large HDL particles | mmol/l |
| L-HDL-L | Total lipids in large HDL | mmol/l |
| L-HDL-PL | Phospholipids in large HDL | mmol/l |
| L-HDL-C | Cholesterol in large HDL | mmol/l |
| L-HDL-CE | Cholesteryl esters in large HDL | mmol/l |
| L-HDL-FC | Free cholesterol in large HDL | mmol/l |
| L-HDL-TG | Triglycerides in large HDL | mmol/l |
| M-HDL-P | Concentration of medium HDL particles | mmol/l |
| M-HDL-L | Total lipids in medium HDL | mmol/l |
| M-HDL-PL | Phospholipids in medium HDL | mmol/l |
| M-HDL-C | Cholesterol in medium HDL | mmol/l |
| M-HDL-CE | Cholesteryl esters in medium HDL | mmol/l |
| M-HDL-FC | Free cholesterol in medium HDL | mmol/l |
| M-HDL-TG | Triglycerides in medium HDL | mmol/l |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 18/28 |

| S-HDL-L Total lipids in small HDL S-HDL-PL S-HDL-CC Cholesterol in small HDL S-HDL-CC Cholesteryl in small HDL S-HDL-CC Cholesteryl in small HDL S-HDL-FC Free cholesterol in small HDL S-HDL-FC Free cholesterol in small HDL S-HDL-FC Triglycerides in small HDL S-HDL-FC Triglycerides in small HDL S-HDL-TG Triglycerides in small HDL SXL-VLDL-CC Cholesterol to total lipids ratio in chylomicrons and extremely large VLDL SXL-VLDL-CC SC Cholesterol to total lipids ratio in chylomicrons and extremely large VLDL SXL-VLDL-TG Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL SXL-VLDL-TG Triglycerides to total lipids ratio in very large VLDL SXL-VLDL-CC Cholesterol to total lipids ratio in very large VLDL SXL-VLDL-CC Cholesterol to total lipids ratio in very large VLDL SXL-VLDL-CC SC Cholesteryl exters to total lipids ratio in very large VLDL SXL-VLDL-TG Triglycerides to total lipids ratio in very large VLDL SXL-VLDL-TG Triglycerides to total lipids ratio in very large VLDL SXL-VLDL-TG Triglycerides to total lipids ratio in very large VLDL SXL-VLDL-TG Triglycerides to total lipids ratio in very large VLDL SC L-VLDL-TG Triglycerides to total lipids ratio in medium VLDL SC L-VLDL-TG Triglycerides to total lipids ratio in medium VLDL SC L-VLDL-TG Triglycerides to total lipids ratio in medium VLDL SC S-VLDL-TG Triglycerides to total lipids ratio in small VLDL SC S-VLDL-TG Triglycerides to total lipids ratio in small VLDL SC S-VLDL-TG Triglycerides to tot | S-HDL-P | Concentration of small HDL particles | mmol/l |
|---|---|---|---|
| S-HDL-PL Phospholipids in small HDL mmol/l S-HDL-C Cholesterol in small HDL mmol/l S-HDL-FC Free cholesterol to total lipids ratio in chylomicrons and extremely large VLDL % XXL-VLDL-PL % Cholesterol to total lipids ratio in chylomicrons and extremely large VLDL % XXL-VLDL-FC % Cholesteryl esters to total lipids ratio in chylomicrons and extremely large VLDL % XXL-VLDL-FC % Free cholesterol to total lipids ratio in chylomicrons and extremely large VLDL % XXL-VLDL-FC % Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL % XXL-VLDL-FC % Cholesterol to total lipids ratio in very large VLDL % XL-VLDL-CE % Cholesterol to total lipids ratio in very large VLDL % XL-VLDL-CE % Cholesterol to total lipids ratio in very large VLDL % XL-VLDL-FC % Prec cholesterol to total lipids ratio in very large VLDL % XL-VLDL-FC % Cholesterol to total lipids ratio in very large VLDL % XL-VLDL-FC % Prec cholesterol to total lipids ratio in very large VLDL % XL-VLDL-FC % Prec cholesterol to total lipids ratio in very large VLDL % XL-VLDL-FC % Prec cholesterol to total lipids ratio in large VLDL % XL-VLDL-FC % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Cholesterol to total lipids ratio in large VLDL % M-VLDL-FC % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Cholesterol to total lipids ratio in medium VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in medium VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in medium | | | |
| S-HDL-C Cholesterol in small HDL S-HDL-CE Cholesteryl esters in small HDL S-HDL-TG Triglycerides in small HDL XXL-VLDL-PL Phospholipids to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-CC Cholesterol to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-CC Cholesterol to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-CC Cholesterol to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-TG Free cholesterol to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-TG Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-TG Triglycerides to total lipids ratio in very large VLDL XXL-VLDL-CC Cholesterol to total lipids ratio in very large VLDL XXL-VLDL-CC Cholesterol to total lipids ratio in very large VLDL XXL-VLDL-CC Cholesterol to total lipids ratio in very large VLDL XXL-VLDL-TG Triglycerides to total lipids ratio in very large VLDL XXL-VLDL-TG Triglycerides to total lipids ratio in very large VLDL XXL-VLDL-TG Triglycerides to total lipids ratio in very large VLDL XXL-VLDL-TG Triglycerides to total lipids ratio in very large VLDL X-VLDL-TG Triglycerides to total lipids ratio in large VLDL X-VLDL-CC Cholesterol to total lipids ratio in large VLDL X-VLDL-CC Cholesterol to total lipids ratio in large VLDL X-VLDL-CC Cholesterol to total lipids ratio in large VLDL X-VLDL-TG Triglycerides to total lipids ratio in medium VLDL X-VLDL-TG Triglycerides to total lipids ratio in medium VLDL X-VLDL-TG Triglycerides to total lipids ratio in medium VLDL X-VLDL-TG Triglycerides to total lipids ratio in medium VLDL X-VLDL-TG Triglycerides to total lip | | | |
| S-HDL-CE Cholesteryl esters in small HDL S-HDL-FC Free cholesterol in small HDL XXL-VLDL-PL Prospholipids to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-CS Cholesterol to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-CS Cholesteryl esters to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-FC Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-FC Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-FC Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-CS Cholesterol to total lipids ratio in very large VLDL XL-VLDL-CS Cholesterol to total lipids ratio in very large VLDL XL-VLDL-FC Triglycerides to total lipids ratio in very large VLDL XL-VLDL-FC Triglycerides to total lipids ratio in very large VLDL XL-VLDL-FC Triglycerides to total lipids ratio in very large VLDL XL-VLDL-FC Cholesterol to total lipids ratio in very large VLDL XL-VLDL-FC Cholesterol to total lipids ratio in very large VLDL XL-VLDL-CS Cholesterol to total lipids ratio in very large VLDL CVLDL-CS Cholesterol to total lipids ratio in large VLDL Cholesterol to total lipids ratio in large VLDL Cholesterol to total lipids ratio in large VLDL Cholesterol to total lipids ratio in large VLDL Cholesterol Serve to total lipids ratio in large VLDL Cholesterol Serve to total lipids ratio in large VLDL Cholesterol Serve total lipids ratio in large VLDL Cholesterol Serve total lipids ratio in large VLDL Cholesterol Serve total lipids ratio in large VLDL Cholesterol Serve total lipids ratio in medium VLDL % N-VLDL-CS Cholesterol Serve to total lipids ratio in medium VLDL % N-VLDL-CS Cholesterol Serve total lipids ratio in medium VLDL % S-VLDL-CS Cholesterol Serve total lipids ratio in small VLDL % S-VLDL-CS Cholesterol Serve total lipids ratio in small VLDL % S-VLDL-CS Cholesterol Serve total lipids ratio in small VLDL % S-VLDL-CS Chol | | | |
| S-HDL-FC Free cholesterol in small HDL Mmol/I XXL-VLDL-PL % Phospholipids to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-CE % Cholesterol to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-CE % Cholesterol to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-FC % Free cholesterol to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-FG % Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-PG % Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-C % Cholesterol to total lipids ratio in very large VLDL XL-VLDL-G % Cholesterol to total lipids ratio in very large VLDL XL-VLDL-FC % Cholesterol to total lipids ratio in very large VLDL XL-VLDL-FG % Triglycerides to total lipids ratio in very large VLDL XL-VLDL-FG % Triglycerides to total lipids ratio in very large VLDL XL-VLDL-FG % Triglycerides to total lipids ratio in large VLDL VLDL-C % Cholesterol to total lipids ratio in large VLDL VLDL-C % Cholesterol to total lipids ratio in large VLDL VLDL-C % Cholesterol to total lipids ratio in large VLDL VLDL-C % Cholesterol to total lipids ratio in large VLDL VLDL-FC % Free cholesterol to total lipids ratio in large VLDL VLDL-FC % Free cholesterol to total lipids ratio in large VLDL VLDL-FC % Free cholesterol to total lipids ratio in large VLDL VLDL-FC % Triglycerides to total lipids ratio in medium VLDL M-VLDL-FG % Triglycerides to total lipids ratio in medium VLDL S-VLDL-FG % Triglycerides to total lipids ratio in medium VLDL M-VLDL-FG % Triglycerides to total lipids ratio in medium VLDL S-VLDL-FG % Triglycerides to total lipids ratio in medium VLDL S-VLDL-FG % Triglycerides to total lipids ratio in small VLDL S-VLDL-FG % Cholesterol to total lipids ratio in small VLDL S-VLDL-FG % Cholesterol to total lipids ratio in small VLDL S-VLDL-FG % Cholesterol to total lipids ratio in small VLDL S-VLDL-FG % Cholesterol to | | | |
| S-HDL-TG XXL-VLDL-PL % Phospholipids to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-CC % Cholesteryl esters to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-CC % Cholesteryl esters to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-FC % Free cholesterol to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-TG % Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-PC % Phospholipids to total lipids ratio in very large VLDL XL-VLDL-CC % Cholesterol to total lipids ratio in very large VLDL XL-VLDL-CC % Cholesterol to total lipids ratio in very large VLDL XL-VLDL-TG % Triglycerides to total lipids ratio in very large VLDL XL-VLDL-TG % Triglycerides to total lipids ratio in very large VLDL XL-VLDL-TG % Triglycerides to total lipids ratio in large VLDL VLDL-CC % Cholesterol to total lipids ratio in large VLDL VLDL-CC % Cholesterol to total lipids ratio in large VLDL VLDL-CC % Cholesterol to total lipids ratio in large VLDL VLDL-CC % Cholesterol to total lipids ratio in large VLDL VLDL-TG % Triglycerides to total lipids ratio in large VLDL VLDL-TG % Triglycerides to total lipids ratio in large VLDL VLDL-TG % Triglycerides to total lipids ratio in large VLDL VLDL-TG % Triglycerides to total lipids ratio in large VLDL VLDL-TG % Triglycerides to total lipids ratio in medium VLDL % VLDL-CC % Cholesterol to total lipids ratio in medium VLDL % VLDL-CC % Cholesterol to total lipids ratio in medium VLDL % VLDL-TG % Triglycerides to total lipids ratio in small VLDL % VLDL-TG % | | | |
| XXL-VLDL-C % Cholesteryl esters to total lipids ratio in chylomicrons and extremely large VLDL % XXL-VLDL-CE % Cholesteryl esters to total lipids ratio in chylomicrons and extremely large VLDL % XXL-VLDL-FC % Free cholesterol to total lipids ratio in chylomicrons and extremely large VLDL % XXL-VLDL-FC % Free cholesterol to total lipids ratio in chylomicrons and extremely large VLDL % XXL-VLDL-TG % Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL % XXL-VLDL-TG % Cholesterol to total lipids ratio in very large VLDL % XL-VLDL-C % Cholesterol to total lipids ratio in very large VLDL % XL-VLDL-C % Cholesterol to total lipids ratio in very large VLDL % XL-VLDL-TG % Triglycerides to total lipids ratio in very large VLDL % XL-VLDL-TG % Free cholesterol to total lipids ratio in very large VLDL % XL-VLDL-TG % Triglycerides to total lipids ratio in very large VLDL % L-VLDL-C % Cholesterol to total lipids ratio in large VLDL % L-VLDL-C % Cholesterol to total lipids ratio in large VLDL % L-VLDL-C % Cholesterol to total lipids ratio in large VLDL % L-VLDL-C % Cholesterol to total lipids ratio in large VLDL % L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % M-VLDL-C % Cholesterol to total lipids ratio in large VLDL % M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL % S-VLDL-C % Cholesterol to total lipids ratio in medium VLDL % S-VLDL-C % Cholesterol to total lipids ratio in medium VLDL % S-VLDL-C % Cholesterol to total lipids ratio in medium VLDL % S-VLDL-C % Cholesterol to total lipids ratio in small VLDL % S-VLDL-C % Cholesterol to total lipids ratio in small VLDL % S-VLDL-C % Cholesterol to total lipids ratio in small VLDL % S-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % S-V | | | |
| XXL-VLDL-CE % Cholesterol to total lipids ratio in chylomicrons and extremely large VLDL % XXL-VLDL-FC % Free cholesterol to total lipids ratio in chylomicrons and extremely large VLDL % XXL-VLDL-FC % Free cholesterol to total lipids ratio in chylomicrons and extremely large VLDL % XXL-VLDL-TG % Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL % XL-VLDL-PL % Phospholipids to total lipids ratio in very large VLDL % XL-VLDL-CE % Cholesterol to total lipids ratio in very large VLDL % XL-VLDL-FC % Triglycerides to total lipids ratio in very large VLDL % XL-VLDL-FC % Triglycerides to total lipids ratio in very large VLDL % XL-VLDL-FC % Triglycerides to total lipids ratio in very large VLDL % XL-VLDL-FC % The cholesterol to total lipids ratio in large VLDL % L-VLDL-CP & Phospholipids to total lipids ratio in large VLDL % L-VLDL-FC % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Triglycerides to total lipids ratio in large VLDL % L-VLDL-FC % Triglycerides to total lipids ratio in large VLDL % M-VLDL-FC % Triglycerides to total lipids ratio in large VLDL % M-VLDL-FC % Triglycerides to total lipids ratio in large VLDL % M-VLDL-FC % Triglycerides to total lipids ratio in medium VLDL % M-VLDL-CP & Cholesterol to total lipids ratio in medium VLDL % M-VLDL-CP & Cholesterol to total lipids ratio in medium VLDL % M-VLDL-CP & Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % S-VLDL-CP & Cholesterol to total lipids ratio in small VLDL % S-VLDL-CP & Phospholipids to total lipids ratio in small VLDL % S-VLDL-CF % Triglycerides to total lipids ratio in small VLDL % S-VLDL-CF % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-CF % Free cholesterol to total lipids ratio in very small VLDL % S-VLDL-CF % Triglycerides to total lipids ratio in very sma | | | |
| XXL-VLDL-CE % Cholesteryl esters to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-FC % Free cholesterol to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-TG % Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL XL-VLDL-PL % Phospholipids to total lipids ratio in very large VLDL XL-VLDL-C % Cholesterol to total lipids ratio in very large VLDL XL-VLDL-FC % Cholesterol to total lipids ratio in very large VLDL XL-VLDL-TG % Free cholesterol to total lipids ratio in very large VLDL XL-VLDL-TG % Triglycerides to total lipids ratio in very large VLDL L-VLDL-C % Cholesterol to total lipids ratio in very large VLDL L-VLDL-C % Cholesterol to total lipids ratio in large VLDL L-VLDL-C % Cholesterol to total lipids ratio in large VLDL L-VLDL-C % Cholesterol to total lipids ratio in large VLDL L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL M-VLDL-TG % Triglycerides to total lipids ratio in large VLDL M-VLDL-C % Cholesterol to total lipids ratio in large VLDL M-VLDL-C % Cholesterol to total lipids ratio in large VLDL M-VLDL-TG % Triglycerides to total lipids ratio in large VLDL M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL M-VLDL-G % Cholesterol to total lipids ratio in medium VLDL M-VLDL-G % Cholesterol to total lipids ratio in medium VLDL M-VLDL-G % Cholesterol to total lipids ratio in small VLDL S-VLDL-C % Cholesterol to total lipids ratio in very small VLDL S-VLDL-C % Cholesterol to total lipids ratio in very small VLDL S-VLDL-C % Cholesterol to total lipids ratio in very small VLDL S-VLD | XXL-VLDL-PL % | Phospholipids to total lipids ratio in chylomicrons and extremely large VLDL | 70 |
| XXL-VLDL-FC % Free cholesterol to total lipids ratio in chylomicrons and extremely large VLDL XXL-VLDL-TG % Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL XL-VLDL-C % Cholesterol to total lipids ratio in very large VLDL XL-VLDL-C % Cholesterol to total lipids ratio in very large VLDL XL-VLDL-FC % Free cholesterol to total lipids ratio in very large VLDL XL-VLDL-TG % Triglycerides to total lipids ratio in very large VLDL XL-VLDL-TG % Triglycerides to total lipids ratio in very large VLDL XL-VLDL-C % Cholesterol to total lipids ratio in very large VLDL L-VLDL-C % Cholesterol to total lipids ratio in large VLDL L-VLDL-C % Cholesterol to total lipids ratio in large VLDL L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL M-VLDL-TG % Triglycerides to total lipids ratio in large VLDL M-VLDL-TG % Triglycerides to total lipids ratio in large VLDL M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL M-VLDL-FC % Triglycerides to total lipids ratio in medium VLDL M-VLDL-FC % Triglycerides to total lipids ratio in medium VLDL M-VLDL-FC % Triglycerides to total lipids ratio in medium VLDL M-VLDL-FC % Triglycerides to total lipids ratio in medium VLDL M-VLDL-FC % Triglycerides to total lipids ratio in small VLDL S-VLDL-C % Cholesterol to total lipids ratio in small VLDL S-VLDL-C % Cholesterol to total lipids ratio in small VLDL S-VLDL-FC % Triglycerides to total lipids ratio in small VLDL S-VLDL-FC % Triglycerides to total lipids ratio in small VLDL S-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL S-VLDL-FC % Cholesterol to total lipids ratio in very small VLDL S-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL S-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL | XXL-VLDL-C % | Cholesterol to total lipids ratio in chylomicrons and extremely large VLDL | % |
| XXL-VLDL-TG % Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL % XL-VLDL-PL % Phospholipids to total lipids ratio in very large VLDL % XL-VLDL-C6 % Cholesterol to total lipids ratio in very large VLDL % XL-VLDL-C7 % Cholesterol esters to total lipids ratio in very large VLDL % XL-VLDL-C7 % Free cholesterol to total lipids ratio in very large VLDL % XL-VLDL-TG % Free cholesterol to total lipids ratio in very large VLDL % XL-VLDL-PC % Phospholipids to total lipids ratio in very large VLDL % L-VLDL-PC % Phospholipids to total lipids ratio in large VLDL % L-VLDL-C6 % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Free cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Free cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Free cholesterol to total lipids ratio in large VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in large VLDL % M-VLDL-FC % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-C7 % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-C8 % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-C7 % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-C8 % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesteryl esters to total lipids ratio in very small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % S-VLDL-FC % Cholesteryl esters to total lipids ratio in very small VLDL % S-VLDL-FC % Free cholesterol to tota | XXL-VLDL-CE % | Cholesteryl esters to total lipids ratio in chylomicrons and extremely large VLDL | % |
| XL-VLDL-PL % Phospholipids to total lipids ratio in very large VLDL % XL-VLDL-CE % Cholesterol to total lipids ratio in very large VLDL % XL-VLDL-PC % Cholesterol esters to total lipids ratio in very large VLDL % XL-VLDL-PC % Free cholesterol to total lipids ratio in very large VLDL % XL-VLDL-PG % Free cholesterol to total lipids ratio in very large VLDL % XL-VLDL-PL % Phospholipids to total lipids ratio in large VLDL % L-VLDL-PC % Cholesterol to total lipids ratio in large VLDL % L-VLDL-PC % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Free cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Free cholesterol to total lipids ratio in large VLDL % M-VLDL-PL % Phospholipids to total lipids ratio in large VLDL % M-VLDL-PC % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-PC % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-CE % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-PC % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-CE % Cholesteryl esters to total lipids ratio in very small VLDL % S-VLDL-CE % Cholesteryl esters to total lipids ratio in very small VLDL % S-VLDL-CE % Cholesteryl esters to total lipids ratio in very small VLDL % S-VLDL-CE % Chol | XXL-VLDL-FC % | Free cholesterol to total lipids ratio in chylomicrons and extremely large VLDL | % |
| XL-VLDL-C % Cholesterol to total lipids ratio in very large VLDL % XL-VLDL-FC % Free cholesterol to total lipids ratio in very large VLDL % XL-VLDL-FC % Free cholesterol to total lipids ratio in very large VLDL % XL-VLDL-TG % Triglycerides to total lipids ratio in very large VLDL % XL-VLDL-PC % Phospholipids to total lipids ratio in large VLDL % L-VLDL-C % Cholesterol to total lipids ratio in large VLDL % L-VLDL-CE % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Triglycerides to total lipids ratio in large VLDL % L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % M-VLDL-PL % Phospholipids to total lipids ratio in large VLDL % M-VLDL-CE % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-CE % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-CE % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Triglycerides to total lipids ratio in medium VLDL % M-VLDL-FC % Triglycerides to total lipids ratio in medium VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in medium VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-PC % Triglycerides to total lipids ratio in small VLDL % S-VLDL-PC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-PC % Triglycerides to total lipids ratio in small VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in very small VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in very small VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in very small VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in very small VLDL % S-VLDL-PC % Free cholesterol to total lipids ratio in very small VLDL % S-VLDL-PC % Free cholesterol to total lipids ratio in very small VLDL % S-VLDL-PC % Free cho | XXL-VLDL-TG % | Triglycerides to total lipids ratio in chylomicrons and extremely large VLDL | % |
| XL-VLDL-C % Cholesterol to total lipids ratio in very large VLDL % XL-VLDL-FC % Free cholesterol to total lipids ratio in very large VLDL % XL-VLDL-FC % Free cholesterol to total lipids ratio in very large VLDL % XL-VLDL-TG % Triglycerides to total lipids ratio in very large VLDL % XL-VLDL-PL % Phospholipids to total lipids ratio in large VLDL % L-VLDL-C % Cholesterol to total lipids ratio in large VLDL % L-VLDL-C % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Triglycerides to total lipids ratio in large VLDL % L-VLDL-FC % Triglycerides to total lipids ratio in large VLDL % M-VLDL-FC % Triglycerides to total lipids ratio in large VLDL % M-VLDL-CE % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-CE % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Triglycerides to total lipids ratio in medium VLDL % M-VLDL-FC % Triglycerides to total lipids ratio in medium VLDL % M-VLDL-FC % Triglycerides to total lipids ratio in medium VLDL % M-VLDL-FC % Triglycerides to total lipids ratio in medium VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in very small VLDL % S-VLDL-FC % Cholesterol total lipids ratio in very small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL % S-VLDL-FC % Triglycerid | XL-VLDL-PL % | Phospholipids to total lipids ratio in very large VLDL | % |
| XL-VLDL-FC % Free cholesterol to total lipids ratio in very large VLDL % XL-VLDL-TG % Triglycerides to total lipids ratio in very large VLDL % L-VLDL-PL % Phospholipids to total lipids ratio in large VLDL % L-VLDL-C % Cholesterol to total lipids ratio in large VLDL % L-VLDL-CE % Cholesteryl esters to total lipids ratio in large VLDL % L-VLDL-TG % Free cholesterol to total lipids ratio in large VLDL % L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % M-VLDL-CE % Cholesterol to total lipids ratio in macdium VLDL % M-VLDL-CF % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-CF % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Triglycerides to total lipids ratio in medium VLDL % M-VLDL-TG % Triglycerides to total lipids ratio in medium VLDL % S-VLDL-PL % Phospholipids to total lipids ratio in small VLDL % S-VLDL-CF % Cholesterol to total lipids ratio in small VLDL % S-VLDL-CF % Cholesterol to total lipids ratio in small VLDL % S-VLDL-CF % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in very small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free choles | XL-VLDL-C % | Cholesterol to total lipids ratio in very large VLDL | % |
| XL-VLDL-FC % Free cholesterol to total lipids ratio in very large VLDL % XL-VLDL-TG % Triglycerides to total lipids ratio in very large VLDL % L-VLDL-PL % Phospholipids to total lipids ratio in large VLDL % L-VLDL-C % Cholesterol to total lipids ratio in large VLDL % L-VLDL-CE % Cholesterol to total lipids ratio in large VLDL % L-VLDL-FC % Free cholesterol to total lipids ratio in large VLDL % L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % M-VLDL-PL % Phospholipids to total lipids ratio in medium VLDL % M-VLDL-CF % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-CF % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % S-VLDL-PL % Phospholipids to total lipids ratio in small VLDL % S-VLDL-PC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-CF % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in very small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS | XL-VLDL-CE % | | % |
| L-VLDL-PL % Phospholipids to total lipids ratio in large VLDL % L-VLDL-C % Cholesterol to total lipids ratio in large VLDL % L-VLDL-CE % Cholesteryl esters to total lipids ratio in large VLDL % L-VLDL-FC % Free cholesterol to total lipids ratio in large VLDL % L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % M-VLDL-PL % Phospholipids to total lipids ratio in medium VLDL % M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-CE % Cholesteryl esters to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-TG % Triglycerides to total lipids ratio in medium VLDL % M-VLDL-TG % Triglycerides to total lipids ratio in medium VLDL % S-VLDL-PL % Phospholipids to total lipids ratio in small VLDL % S-VLDL-C % Cholesterol to total lipids ratio in small VLDL % S-VLDL-CE % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Triglycerides to total lipids ratio in small VLDL % S-VLDL-FC % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Cholesteryl esters to total lipids ratio in very small VLDL % XS-VLDL-FC % Cholesteryl esters to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Phospholipids to total lipids ratio in very small VLDL % | XL-VLDL-FC % | | % |
| L-VLDL-C % Cholesterol to total lipids ratio in large VLDL % L-VLDL-CE % Cholesteryl esters to total lipids ratio in large VLDL % L-VLDL-FC % Free cholesterol to total lipids ratio in large VLDL % L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % M-VLDL-PL % Phospholipids to total lipids ratio in medium VLDL % M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-CE % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % S-VLDL-PL % Phospholipids to total lipids ratio in small VLDL % S-VLDL-CE % Cholesterol to total lipids ratio in small VLDL % S-VLDL-CE % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-FC % Phospholipids to total lipids ratio in very small VLDL % | XL-VLDL-TG % | Triglycerides to total lipids ratio in very large VLDL | % |
| L-VLDL-CE % Cholesteryl esters to total lipids ratio in large VLDL % L-VLDL-FC % Free cholesterol to total lipids ratio in large VLDL % L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % M-VLDL-PL % Phospholipids to total lipids ratio in medium VLDL % M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-CE % Cholesteryl esters to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-FG % Free cholesterol to total lipids ratio in medium VLDL % S-VLDL-PL % Phospholipids to total lipids ratio in small VLDL % S-VLDL-CE % Cholesterol to total lipids ratio in small VLDL % S-VLDL-CE % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-FC % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-FC % Phospholipids to total lipids ratio in very small VLDL % | L-VLDL-PL % | Phospholipids to total lipids ratio in large VLDL | % |
| L-VLDL-FC % Free cholesterol to total lipids ratio in large VLDL % L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % M-VLDL-PL % Phospholipids to total lipids ratio in medium VLDL % M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-CE % Cholesteryl esters to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-TG % Triglycerides to total lipids ratio in medium VLDL % S-VLDL-PL % Phospholipids to total lipids ratio in small VLDL % S-VLDL-C % Cholesterol to total lipids ratio in small VLDL % S-VLDL-CE % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % S-VLDL-TG % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-TG % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-TG % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-TG % Phospholipids to total lipids ratio in very small VLDL % | L-VLDL-C % | Cholesterol to total lipids ratio in large VLDL | % |
| L-VLDL-TG % Triglycerides to total lipids ratio in large VLDL % M-VLDL-PL % Phospholipids to total lipids ratio in medium VLDL % M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Cholesteryl esters to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-TG % Triglycerides to total lipids ratio in medium VLDL % S-VLDL-PL % Phospholipids to total lipids ratio in small VLDL % S-VLDL-C % Cholesterol to total lipids ratio in small VLDL % S-VLDL-C % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % S-VLDL-TG % Cholesterol to total lipids ratio in small VLDL % XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Phospholipids to total lipids ratio in IDL % | L-VLDL-CE % | Cholesteryl esters to total lipids ratio in large VLDL | % |
| M-VLDL-PL % Phospholipids to total lipids ratio in medium VLDL % M-VLDL-CE % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-FC % Cholesteryl esters to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-TG % Triglycerides to total lipids ratio in medium VLDL % S-VLDL-PL % Phospholipids to total lipids ratio in small VLDL % S-VLDL-C % Cholesterol to total lipids ratio in small VLDL % S-VLDL-CE % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % S-VLDL-TG % Cholesterol to total lipids ratio in small VLDL % XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-TG % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-TG % Phospholipids to total lipids ratio in very small VLDL % | L-VLDL-FC % | Free cholesterol to total lipids ratio in large VLDL | % |
| M-VLDL-C % Cholesterol to total lipids ratio in medium VLDL % M-VLDL-CE % Cholesteryl esters to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-TG % Triglycerides to total lipids ratio in medium VLDL % S-VLDL-PL % Phospholipids to total lipids ratio in small VLDL % S-VLDL-C % Cholesterol to total lipids ratio in small VLDL % S-VLDL-CE % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Tree cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % DL-PL % Phospholipids to total lipids ratio in IDL % | L-VLDL-TG % | Triglycerides to total lipids ratio in large VLDL | % |
| M-VLDL-CE % Cholesteryl esters to total lipids ratio in medium VLDL % M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % S-VLDL-PL % Phospholipids to total lipids ratio in small VLDL % S-VLDL-C % Cholesterol to total lipids ratio in small VLDL % S-VLDL-FC % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesteryl esters to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % DL-PL % Phospholipids to total lipids ratio in IDL % | M-VLDL-PL % | Phospholipids to total lipids ratio in medium VLDL | % |
| M-VLDL-FC % Free cholesterol to total lipids ratio in medium VLDL % M-VLDL-TG % Triglycerides to total lipids ratio in medium VLDL % S-VLDL-PL % Phospholipids to total lipids ratio in small VLDL % S-VLDL-C % Cholesterol to total lipids ratio in small VLDL % S-VLDL-CE % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % DL-PL % Phospholipids to total lipids ratio in IDL % | M-VLDL-C % | Cholesterol to total lipids ratio in medium VLDL | % |
| M-VLDL-TG % Triglycerides to total lipids ratio in medium VLDL % S-VLDL-PL % Phospholipids to total lipids ratio in small VLDL % S-VLDL-C % Cholesterol to total lipids ratio in small VLDL % S-VLDL-CE % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesteryl esters to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Phospholipids to total lipids ratio in very small VLDL % IDL-PL % Phospholipids to total lipids ratio in IDL % | M-VLDL-CE % | Cholesteryl esters to total lipids ratio in medium VLDL | % |
| S-VLDL-PL % Phospholipids to total lipids ratio in small VLDL % S-VLDL-C % Cholesterol to total lipids ratio in small VLDL % S-VLDL-CE % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesteryl esters to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % DL-PL % Phospholipids to total lipids ratio in IDL % | M-VLDL-FC % | Free cholesterol to total lipids ratio in medium VLDL | % |
| S-VLDL-C % Cholesterol to total lipids ratio in small VLDL % S-VLDL-CE % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesteryl esters to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % IDL-PL % Phospholipids to total lipids ratio in IDL % | M-VLDL-TG % | Triglycerides to total lipids ratio in medium VLDL | % |
| S-VLDL-CE % Cholesteryl esters to total lipids ratio in small VLDL % S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesteryl esters to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % XS-VLDL-TG % Phospholipids to total lipids ratio in IDL % | S-VLDL-PL % | Phospholipids to total lipids ratio in small VLDL | % |
| S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesteryl esters to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % IDL-PL % Phospholipids to total lipids ratio in IDL % | S-VLDL-C % | Cholesterol to total lipids ratio in small VLDL | % |
| S-VLDL-FC % Free cholesterol to total lipids ratio in small VLDL % S-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesteryl esters to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % IDL-PL % Phospholipids to total lipids ratio in IDL % | | Cholesteryl esters to total lipids ratio in small VLDL | % |
| S-VLDL-TG % Triglycerides to total lipids ratio in small VLDL % XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesteryl esters to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % IDL-PL % Phospholipids to total lipids ratio in IDL % | | | % |
| XS-VLDL-PL % Phospholipids to total lipids ratio in very small VLDL % XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesteryl esters to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % IDL-PL % Phospholipids to total lipids ratio in IDL % | | | |
| XS-VLDL-C % Cholesterol to total lipids ratio in very small VLDL % XS-VLDL-CE % Cholesteryl esters to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % IDL-PL % Phospholipids to total lipids ratio in IDL % | | | % |
| XS-VLDL-CE % Cholesteryl esters to total lipids ratio in very small VLDL % XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % IDL-PL % Phospholipids to total lipids ratio in IDL % | | | % |
| XS-VLDL-FC % Free cholesterol to total lipids ratio in very small VLDL % XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % IDL-PL % Phospholipids to total lipids ratio in IDL % | | | |
| XS-VLDL-TG % Triglycerides to total lipids ratio in very small VLDL % IDL-PL % Phospholipids to total lipids ratio in IDL % | | | |
| IDL-PL % Phospholipids to total lipids ratio in IDL % | | | |
| | IDL-C % | | % |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 19/28 |

| IDL-CE % | Cholesteryl esters to total lipids ratio in IDL | % |
|-------------|------------------------------------------------------------|---|
| IDL-FC % | Free cholesterol to total lipids ratio in IDL | % |
| IDL-TG % | Triglycerides to total lipids ratio in IDL | % |
| L-LDL-PL % | Phospholipids to total lipids ratio in large LDL | % |
| L-LDL-C % | Cholesterol to total lipids ratio in large LDL | % |
| L-LDL-CE % | Cholesteryl esters to total lipids ratio in large LDL | % |
| L-LDL-FC % | Free cholesterol to total lipids ratio in large LDL | % |
| L-LDL-TG % | Triglycerides to total lipids ratio in large LDL | % |
| M-LDL-PL % | Phospholipids to total lipids ratio in medium LDL | % |
| M-LDL-C % | Cholesterol to total lipids ratio in medium LDL | % |
| M-LDL-CE % | Cholesteryl esters to total lipids ratio in medium LDL | % |
| M-LDL-FC % | Free cholesterol to total lipids ratio in medium LDL | % |
| M-LDL-TG % | Triglycerides to total lipids ratio in medium LDL | % |
| S-LDL-PL % | Phospholipids to total lipids ratio in small LDL | % |
| S-LDL-C % | Cholesterol to total lipids ratio in small LDL | % |
| S-LDL-CE % | Cholesteryl esters to total lipids ratio in small LDL | % |
| S-LDL-FC % | Free cholesterol to total lipids ratio in small LDL | % |
| S-LDL-TG % | Triglycerides to total lipids ratio in small LDL | % |
| XL-HDL-PL % | Phospholipids to total lipids ratio in very large HDL | % |
| XL-HDL-C % | Cholesterol to total lipids ratio in very large HDL | % |
| XL-HDL-CE % | Cholesteryl esters to total lipids ratio in very large HDL | % |
| XL-HDL-FC % | Free cholesterol to total lipids ratio in very large HDL | % |
| XL-HDL-TG % | Triglycerides to total lipids ratio in very large HDL | % |
| L-HDL-PL % | Phospholipids to total lipids ratio in large HDL | % |
| L-HDL-C % | Cholesterol to total lipids ratio in large HDL | % |
| L-HDL-CE % | Cholesteryl esters to total lipids ratio in large HDL | % |
| L-HDL-FC % | Free cholesterol to total lipids ratio in large HDL | % |
| L-HDL-TG % | Triglycerides to total lipids ratio in large HDL | % |
| M-HDL-PL % | Phospholipids to total lipids ratio in medium HDL | % |
| M-HDL-C % | Cholesterol to total lipids ratio in medium HDL | % |
| M-HDL-CE % | Cholesteryl esters to total lipids ratio in medium HDL | % |
| M-HDL-FC % | Free cholesterol to total lipids ratio in medium HDL | % |
| M-HDL-TG % | Triglycerides to total lipids ratio in medium HDL | % |
| S-HDL-PL % | Phospholipids to total lipids ratio in small HDL | % |
| S-HDL-C % | Cholesterol to total lipids ratio in small HDL | % |
| S-HDL-CE % | Cholesteryl esters to total lipids ratio in small HDL | % |
| S-HDL-FC % | Free cholesterol to total lipids ratio in small HDL | % |
| S-HDL-TG % | Triglycerides to total lipids ratio in small HDL | % |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 20/28 |

Table 4: Comparative Analysis of Metabolomic Pre-test and Post-test Results for Placebo Group Blood Samples

| Significance(p-value) | Feature | Mean(after) | Mean(before) | Method | FC | Log2(FC) | -Log10(p-value) | -Log10(padj) |
|---|---|---|---|---|---|---|---|---|
| ves | Creatinine | 64.21 | | | 0.923 | -0.115 | 2.023 | 0.103 |
| yes | IDL CE pct | 51.149 | | | 0.97 | -0.044 | 2.623 | 0.527 |
| yes | IDL C pct | 67.73 | | | 0.976 | -0.035 | 2.767 | 0.527 |
| yes | IDL TG pct | 8.787 | | | 1.147 | 0.197 | 1.332 | 0.06 |
| yes | L LDL CE pct | 53.99 | | | 0.99 | -0.014 | 1.562 | 0.06 |
| yes | L LDL C pct | 71.967 | | | 0.988 | -0.017 | 1.59 | 0.06 |
| yes | L_LDL_TG_pct | 5.966 | | t-test | 1.145 | 0.195 | 1.397 | 0.06 |
| yes | M LDL PL pct | 26.658 | | | 0.987 | -0.019 | 1.452 | 0.06 |
| no | Acetate | 0.017 | | t-test | 1.092 | 0.126 | 0.309 | 0.06 |
| no | Acetoacetate | 0.025 | | t-test | 0.741 | -0.432 | 0.366 | 0.06 |
| no | Acetone | 0.019 | | t-test | 1.063 | 0.089 | 0.067 | 0.005 |
| no | Ala | 0.337 | | t-test | 1.137 | 0.185 | 1.234 | 0.06 |
| no | Albumin | 41.434 | | | 0.98 | -0.029 | 0.259 | 0.06 |
| no | ApoA1 | 1.416 | | t-test | 0.955 | -0.066 | 0.477 | 0.06 |
| no | АроВ | 0.878 | | t-test | 0.977 | -0.033 | 0.24 | 0.06 |
| no | ApoB_by_ApoA1 | 0.63 | | t-test | 1.019 | 0.033 | 0.179 | 0.027 |
| no | bOHbutyrate | 0.094 | | t-test | 1.013 | 0.027 | 0.063 | 0.005 |
| no | Cholines | 2.554 | | t-test | 0.961 | -0.058 | 0.361 | 0.06 |
| no | Citrate | 0.06 | | t-test | 1.043 | 0.050 | 1.126 | 0.06 |
| no | Clinical LDL C | 2.787 | | t-test | 0.933 | -0.101 | 0.605 | 0.06 |
| no | DHA | 0.323 | | t-test | 0.555 | -0.152 | 0.271 | 0.06 |
| no | DHA pct | 2.574 | | t-test | 0.927 | -0.132 | 0.292 | 0.06 |
| no | Gln | 0.487 | | t-test | 1.016 | 0.022 | 0.099 | 0.005 |
| no | Glucose | 4.525 | | t-test | 0.883 | -0.18 | 0.749 | 0.003 |
| no | Gly | 0.251 | | t-test | 1.202 | 0.265 | 1.129 | 0.06 |
| no | GlycA | 0.231 | | t-test | 0.968 | -0.046 | 0.294 | 0.06 |
| no | Glycerol | 0.106 | | t-test | 1.149 | 0.040 | 0.283 | 0.06 |
| no | HDL C | 1.273 | | t-test | 0.93 | -0.105 | 0.283 | 0.06 |
| no | HDL_C | 1.006 | | t-test | 0.935 | -0.103 | 0.733 | 0.06 |
| no | HDL_CE | 0.267 | | t-test | 0.925 | -0.113 | 0.401 | 0.06 |
| no | HDL L | 2.818 | | t-test | 0.947 | -0.077 | 0.461 | 0.06 |
| no | HDL P | 0.016 | | t-test | 0.945 | -0.079 | 0.400 | 0.06 |
| no | HDL PL | 1.426 | | t-test | 0.943 | -0.081 | 0.403 | 0.06 |
| no | HDL_PL | 9.47 | | t-test | 0.931 | -0.072 | 0.403 | 0.00 |
| | | 0.119 | | | 1.082 | 0.113 | 0.142 | 0.01 |
| no | HDL_TG | 0.119 | | t-test | | 0.113 | 0.309 | 0.005 |
| no | His | | | t-test | 1.014 | | | |
| no | IDL_C | 0.779 | | t-test | 0.932 | -0.101 | 0.697 | 0.06 |
| no | IDL_CE | 0.588 | | t-test | 0.925 | -0.112 | 0.755 | 0.06 |
| no | IDL_FC | 0.191 | | t-test | 0.954 | -0.068 | 0.432 | 0.06 |
| no | IDL_FC_pct | 16.581 | | t-test | 0.995 | -0.007 | 0.103 | 0.005 |
| no | IDL_L | 1.143 | | t-test | 0.957 | -0.063 | 0.413 | 0.06 |
| no | IDL_P | 0.269 | | t-test | 0.959 | -0.06 | 0.51 | 0.06 |
| no | IDL_PL | 0.268 | | t-test | 0.973 | -0.039 | 0.233 | 0.06 |
| no | IDL_PL_pct | 23.483 | 23.804 | τ-test | 1.014 | 0.02 | 0.531 | 0.06 |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 21/28 |

| no | IDL TG | 0.095 | 0.106 | t_tost | 1.116 | 0.159 | 0.904 | 0.06 |
|---|---|---|---|---|---|---|---|---|
| no | lle | 0.058 | | t-test | 1.116 | 0.159 | 0.728 | 0.06 |
| no | LA | 4.198 | 4.005 | | 0.954 | -0.068 | 0.447 | 0.06 |
| no | Lactate | 2.987 | 4.773 | | 1.598 | 0.676 | 0.666 | 0.06 |
| no | LA_pct | 33.798 | 33.094 | | 0.979 | -0.03 | 0.269 | 0.06 |
| no | LDL C | 1.974 | 1.859 | | 0.942 | -0.087 | 0.562 | 0.06 |
| no | LDL CE | 1.458 | 1.378 | | 0.945 | -0.082 | 0.526 | 0.06 |
| no | LDL FC | 0.516 | 0.481 | | 0.932 | -0.102 | 0.64 | 0.06 |
| no | LDL L | 2.805 | 2.671 | | 0.952 | -0.102 | 0.455 | 0.06 |
| no | LDL_C | 0.001 | 0.001 | | 0.932 | -0.034 | 0.233 | 0.06 |
| no | LDL_PL | 0.679 | 0.646 | | 0.952 | -0.034 | 0.489 | 0.06 |
| no | LDL_size | 23.873 | 23.877 | | 0.932 | -0.072 | 0.485 | 0.005 |
| | LDL_Size | 0.151 | 0.166 | | 1.097 | 0.133 | 0.715 | 0.003 |
| no | Leu | 0.131 | 0.100 | | 1.145 | 0.133 | 0.713 | 0.06 |
| no | L HDL C | 0.128 | | | 0.884 | -0.178 | 0.729 | |
| no | | | 0.186 | | | | 0.729 | 0.06 |
| no | L_HDL_CE | 0.168 | 0.147 | | 0.876 | -0.191 | | 0.06 |
| no | L_HDL_CE_pct | 35.405 | 31.348 | | 0.885 | -0.176 | 0.669 | 0.06 |
| no | L_HDL_C_pct | 43.805 | 39.532 | | 0.902 | -0.148 | 0.641 | 0.06 |
| no | L_HDL_FC | 0.043 | 0.039 | | 0.916 | -0.126 | 0.386 | 0.06 |
| no | L_HDL_FC_pct | 8.4 | 8.184 | | 0.974 | -0.038 | 0.283 | 0.06 |
| no | L_HDL_L | 0.46 | 0.416 | | 0.905 | -0.144 | 0.532 | 0.06 |
| no | L_HDL_P | 0.001 | 0.001 | | 0.894 | -0.162 | 0.631 | 0.06 |
| no | L_HDL_PL | 0.231 | | t-test | 0.908 | -0.139 | 0.448 | 0.06 |
| no | L_HDL_PL_pct | 51.036 | 52.628 | | 1.031 | 0.044 | 0.609 | 0.06 |
| no | L_HDL_TG | 0.018 | | t-test | 1.111 | 0.151 | 0.24 | 0.06 |
| no | L_HDL_TG_pct | 5.159 | 7.841 | | 1.52 | 0.604 | 0.624 | 0.06 |
| no | L_LDL_C | 1.258 | 1.172 | | 0.932 | -0.101 | 0.64 | 0.06 |
| no | L_LDL_CE | 0.943 | | t-test | 0.933 | -0.1 | 0.626 | 0.06 |
| no | L_LDL_FC | 0.315 | 0.292 | | 0.928 | -0.107 | 0.664 | 0.06 |
| no | L_LDL_FC_pct | 17.977 | 17.673 | | 0.983 | -0.025 | 0.641 | 0.06 |
| no | L_LDL_L | 1.74 | 1.644 | | 0.945 | -0.082 | 0.515 | 0.06 |
| no | L_LDL_P | 0.001 | 0.001 | | 0.978 | -0.032 | 0.192 | 0.032 |
| no | L_LDL_PL | 0.383 | 0.362 | | 0.946 | -0.08 | 0.535 | 0.06 |
| no | L_LDL_PL_pct | 22.067 | 22.033 | | 0.998 | -0.002 | 0.105 | 0.005 |
| no | L_LDL_TG | 0.099 | 0.109 | | 1.103 | 0.142 | 0.794 | 0.06 |
| no | L_VLDL_C | 0.102 | 0.103 | | 1.004 | 0.006 | 0.018 | 0.002 |
| no | L_VLDL_CE | 0.052 | 0.052 | | 0.999 | -0.002 | 0.006 | 0.002 |
| no | L_VLDL_CE_pct | 14.148 | 14.396 | | 1.017 | 0.025 | 0.091 | 0.005 |
| no | L_VLDL_C_pct | 27.766 | 28.219 | | 1.016 | 0.023 | 0.13 | 0.007 |
| no | L_VLDL_FC | 0.05 | 0.051 | | 1.01 | 0.015 | 0.038 | 0.002 |
| no | L_VLDL_FC_pct | 13.618 | 13.824 | | 1.015 | 0.022 | 0.252 | 0.06 |
| no | L_VLDL_L | 0.37 | 0.368 | | 0.994 | -0.008 | 0.018 | 0.002 |
| no | L_VLDL_P | 0 | | t-test | 1.014 | 0.021 | 0.049 | 0.005 |
| no | L_VLDL_PL | 0.072 | 0.074 | | 1.029 | 0.042 | 0.106 | 0.005 |
| no | L_VLDL_PL_pct | 19.037 | 20.007 | | 1.051 | 0.072 | 1.254 | 0.06 |
| no | L_VLDL_TG | 0.195 | 0.191 | | 0.976 | -0.035 | 0.068 | 0.005 |
| no | L_VLDL_TG_pct | 53.196 | 51.774 | | 0.973 | -0.039 | 0.373 | 0.06 |
| no | M_HDL_C | 0.496 | 0.457 | | 0.923 | -0.116 | 0.589 | 0.06 |
| no | M_HDL_CE | 0.412 | 0.381 | | 0.924 | -0.114 | 0.607 | 0.06 |
| no | M_HDL_CE_pct | 41.205 | 40.496 | | 0.983 | -0.025 | 0.385 | 0.06 |
| no | M_HDL_C_pct | 49.479 | 48.641 | | 0.983 | -0.025 | 0.458 | 0.06 |
| no | M_HDL_FC | 0.083 | 0.076 | | 0.917 | -0.124 | 0.497 | 0.06 |
| no | M_HDL_FC_pct | 8.274 | 8.145 | | 0.984 | -0.023 | 0.641 | 0.06 |
| no | M_HDL_L | 0.997 | 0.936 | | 0.939 | -0.09 | 0.444 | 0.06 |
| no | M_HDL_P | 0.004 | 0.003 | | 0.932 | -0.102 | 0.493 | 0.06 |
| no | M_HDL_PL | 0.46 | 0.434 | | 0.944 | -0.082 | 0.399 | 0.06 |
| no | M_HDL_PL_pct | 46.155 | 46.412 | | 1.006 | 0.008 | 0.335 | 0.06 |
| no | M_HDL_TG | 0.042 | 0.045 | | 1.079 | 0.109 | 0.259 | 0.06 |
| no | M_HDL_TG_pct | 4.365 | 4.947 | | 1.133 | 0.181 | 0.511 | 0.06 |
| no | M_LDL_C | 0.507 | 0.485 | | 0.957 | -0.064 | 0.408 | 0.06 |
| no | M_LDL_CE | 0.364 | 0.351 | | 0.965 | -0.052 | 0.326 | 0.06 |
| no | M LDL CE pct | 49.044 | 49.36 | t-test | 1.006 | 0.009 | 0.369 | 0.06 |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 22/28 |

| no | M_LDL_C_pct | 68.369 | 68.131 | t-test | 0.997 | -0.005 | 0.276 | 0.06 |
|---|---|---|---|---|---|---|---|---|
| no | M LDL FC | 0.142 | | t-test | 0.935 | -0.097 | 0.578 | 0.06 |
| no | M_LDL_FC_pct | 19.325 | 18.771 | t-test | 0.971 | -0.042 | 0.947 | 0.06 |
| no | M_LDL_L | 0.739 | 0.71 | t-test | 0.962 | -0.056 | 0.352 | 0.06 |
| no | M_LDL_P | 0 | 0 | t-test | 0.973 | -0.039 | 0.252 | 0.06 |
| no | M LDL PL | 0.196 | 0.187 | t-test | 0.951 | -0.073 | 0.454 | 0.06 |
| no | M_LDL_TG | 0.036 | 0.039 | t-test | 1.094 | 0.129 | 0.657 | 0.06 |
| no | M LDL TG pct | 4.974 | | t-test | 1.118 | 0.161 | 1.087 | 0.06 |
| no | MUFA | 2.749 | | t-test | 0.985 | -0.022 | 0.086 | 0.005 |
| no | MUFA pct | 22.162 | 22.357 | | 1.009 | 0.013 | 0.179 | 0.027 |
| no | M VLDL C | 0.169 | | t-test | 0.946 | -0.081 | 0.334 | 0.06 |
| no | M VLDL CE | 0.088 | | t-test | 0.927 | -0.109 | 0.336 | 0.06 |
| no | M VLDL CE pct | 13.828 | 13.571 | | 0.981 | -0.027 | 0.062 | 0.005 |
| no | M VLDL C pct | 26.337 | 26.195 | | 0.995 | -0.008 | 0.024 | 0.002 |
| no | M VLDL FC | 0.08 | | t-test | 0.966 | -0.05 | 0.255 | 0.06 |
| no | M VLDL FC pct | 12.509 | 12.624 | | 1.009 | 0.013 | 0.078 | 0.005 |
| no | M VLDL L | 0.632 | | t-test | 0.972 | -0.042 | 0.199 | 0.037 |
| no | M VLDL P | 0.032 | | t-test | 0.971 | -0.043 | 0.224 | 0.057 |
| no | M VLDL PL | 0.136 | | t-test | 0.967 | -0.043 | 0.238 | 0.037 |
| no | M VLDL PL pct | 21.162 | 21.384 | | 1.01 | 0.015 | 0.12 | 0.005 |
| | M VLDL TG | 0.327 | | t-test | 0.987 | -0.019 | 0.056 | 0.005 |
| no<br>no | M VLDL_IG M VLDL TG pct | 52.501 | 52.421 | | 0.987 | -0.019 | 0.056 | 0.005 |
| | | 3.425 | | | | -0.002 | 0.482 | |
| no | non_HDL_C | | | t-test | 0.951 | -0.072 | | 0.06<br>0.043 |
| no | Omega_3 | 0.699 | | t-test | 0.901 | | 0.208 | |
| no | Omega_3_pct | 5.426 | | t-test | 0.941 | -0.088 | 0.177 | 0.027 |
| no | Omega_6 | 5.057 | | t-test | 0.955 | -0.066 | 0.533 | 0.06 |
| no | Omega_6_by_Omega_3 | 8.451 | | t-test | 0.982 | -0.026 | 0.063 | 0.005 |
| no | Omega_6_pct | 41.033 | 40.101 | | 0.977 | -0.033 | 0.346 | 0.06 |
| no | Phe | 0.079 | | t-test | 1.073 | 0.102 | 0.361 | 0.06 |
| no | Phosphatidylc | 2.072 | | t-test | 0.966 | -0.049 | 0.262 | 0.06 |
| no | Phosphoglyc | 2.257 | | t-test | 0.961 | -0.058 | 0.303 | 0.06 |
| no | PUFA | 5.756 | | t-test | 0.949 | -0.076 | 0.463 | 0.06 |
| no | PUFA_by_MUFA | 2.103 | | t-test | 0.964 | -0.052 | 0.524 | 0.06 |
| no | PUFA_pct | 46.459 | 45.205 | | 0.973 | -0.039 | 0.775 | 0.06 |
| no | Pyruvate | 0.03 | | t-test | 1.306 | 0.386 | 0.344 | 0.06 |
| no | Remnant_C | 1.451 | 1.4 | t-test | 0.965 | -0.052 | 0.325 | 0.06 |
| no | SFA | 3.901 | | t-test | 1.007 | 0.01 | 0.037 | 0.002 |
| no | SFA_pct | 31.378 | 32.438 | t-test | 1.034 | 0.048 | 0.929 | 0.06 |
| no | S_HDL_C | 0.509 | 0.484 | t-test | 0.95 | -0.074 | 0.56 | 0.06 |
| no | S_HDL_CE | 0.384 | 0.362 | t-test | 0.943 | -0.084 | 0.672 | 0.06 |
| no | S_HDL_CE_pct | 30.584 | 29.951 | t-test | 0.979 | -0.03 | 0.575 | 0.06 |
| no | S_HDL_C_pct | 40.537 | 40.025 | t-test | 0.987 | -0.018 | 0.464 | 0.06 |
| no | S_HDL_FC | 0.125 | 0.121 | t-test | 0.972 | -0.041 | 0.241 | 0.06 |
| no | S_HDL_FC_pct | 9.953 | 10.074 | t-test | 1.012 | 0.017 | 0.587 | 0.06 |
| no | S_HDL_L | 1.256 | 1.209 | t-test | 0.963 | -0.055 | 0.4 | 0.06 |
| no | S_HDL_P | 0.011 | 0.01 | t-test | 0.954 | -0.068 | 0.544 | 0.06 |
| no | S_HDL_PL | 0.694 | 0.669 | t-test | 0.964 | -0.053 | 0.379 | 0.06 |
| no | S_HDL_PL_pct | 55.223 | 55.293 | t-test | 1.001 | 0.002 | 0.078 | 0.005 |
| no | S_HDL_TG | 0.053 | 0.057 | t-test | 1.072 | 0.101 | 0.426 | 0.06 |
| no | S_HDL_TG_pct | 4.24 | 4.682 | t-test | 1.104 | 0.143 | 0.728 | 0.06 |
| no | S LDL C | 0.21 | | t-test | 0.962 | -0.056 | 0.387 | 0.06 |
| no | S LDL CE | 0.15 | | t-test | 0.97 | -0.044 | 0.278 | 0.06 |
| no | S_LDL_CE_pct | 46.01 | | t-test | 1.003 | 0.005 | 0.122 | 0.005 |
| no | S_LDL_C_pct | 64.221 | | t-test | 0.993 | -0.01 | 0.49 | 0.06 |
| no | S LDL FC | 0.059 | | t-test | 0.941 | -0.088 | 0.649 | 0.06 |
| no | S_LDL_FC_pct | 18.211 | | t-test | 0.966 | -0.05 | 0.88 | 0.06 |
| no | S LDL L | 0.326 | | t-test | 0.971 | -0.043 | 0.317 | 0.06 |
| no | S LDL P | 0.520 | | t-test | 0.977 | -0.034 | 0.237 | 0.06 |
| no | S_LDL_PL | 0.1 | | t-test | 0.974 | -0.034 | 0.324 | 0.06 |
| no | S_LDL_PL_pct | 30.746 | | t-test | 0.999 | -0.001 | 0.026 | 0.002 |
| no | S_LDL_TG | 0.016 | | t-test | 1.063 | 0.088 | 0.325 | 0.002 |
| no | S LDL TG pct | 5.032 | | t-test | 1.003 | 0.134 | 0.61 | 0.06 |
| no | Sphingomyelins | 0.448 | | t-test | 0.957 | -0.064 | 0.433 | 0.06 |
| IIU | philligolliae illig | U.440 | 0.428 | i-iest | 0.537 | -0.004 | 0.433 | 0.06 |
| no | S VLDL C | 0.159 | 0.163 | t-test | 1.019 | 0.028 | 0.127 | 0.006 |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 23/28 |

| no | S_VLDL_CE_pct | 21.678 | 22.506 t-test | 1.038 | 0.054 | 0.325 | 0.06 |
|---|---|---|---|---|---|---|---|
| no | S VLDL C pct | 35.59 | 36.258 t-test | 1.019 | 0.027 | 0.146 | 0.01 |
| no | S VLDL FC | 0.062 | 0.061 t-test | 0.985 | -0.022 | 0.101 | 0.005 |
| no | S VLDL FC pct | 13.911 | 13.752 t-test | 0.989 | -0.017 | 0.086 | 0.005 |
| no | S VLDL L | 0.452 | 0.456 t-test | 1.008 | 0.012 | 0.051 | 0.005 |
| no | S VLDL P | 0 | 0 t-test | 1.011 | 0.016 | 0.073 | 0.005 |
| no | S_VLDL_PL | 0.106 | 0.106 t-test | 0.995 | -0.008 | 0.035 | 0.002 |
| no | S_VLDL_PL_pct | 23.642 | 23.475 t-test | 0.993 | -0.01 | 0.095 | 0.005 |
| no | S_VLDL_TG | 0.186 | 0.188 t-test | 1.006 | 0.009 | 0.024 | 0.002 |
| no | S_VLDL_TG_pct | 40.768 | 40.267 t-test | 0.988 | -0.018 | 0.076 | 0.005 |
| no | TG_by_PG | 0.592 | 0.63 t-test | 1.064 | 0.089 | 0.267 | 0.06 |
| no | Total_BCAA | 0.431 | 0.479 t-test | 1.111 | 0.152 | 0.524 | 0.06 |
| no | Total_C | 4.698 | 4.442 t-test | 0.946 | -0.081 | 0.59 | 0.06 |
| no | Total CE | 3.445 | 3.242 t-test | 0.941 | -0.088 | 0.625 | 0.06 |
| no | Total FA | 12.405 | 12.095 t-test | 0.975 | -0.037 | 0.175 | 0.027 |
| no | Total FC | 1.253 | 1.2 t-test | 0.958 | -0.062 | 0.473 | 0.06 |
| no | Total_L | 8.87 | 8.54 t-test | 0.963 | -0.055 | 0.394 | 0.06 |
| | Total P | 0.018 | 0.017 t-test | 0.948 | -0.033 | 0.562 | 0.06 |
| no | | 2.834 | | 0.948 | -0.054 | 0.386 | |
| no | Total_PL | | 2.73 t-test | | | | 0.00 |
| no | Total_TG | 1.338 | 1.367 t-test | 1.022 | 0.031 | 0.078 | 0.005 |
| no | Tyr | 0.055<br>1.44 | 0.061 t-test | 1.109 | 0.15 | 0.463 | 0.06 |
| no | Unsaturation | | 1.407 t-test | 0.977 | -0.033 | 0.814 | 0.06 |
| no | Val | 0.245 | 0.263 t-test | 1.073 | 0.101 | 0.39 | 0.06 |
| no | VLDL_C | 0.672 | 0.674 t-test | 1.003 | 0.004 | 0.016 | 0.002 |
| no | VLDL_CE | 0.394 | 0.396 t-test | 1.004 | 0.005 | 0.021 | 0.002 |
| no | VLDL_FC | 0.278 | 0.278 t-test | 1.001 | 0.002 | 0.008 | 0.002 |
| no | VLDL_L | 2.106 | 2.107 t-test | 1.001 | 0.001 | 0.003 | 0.002 |
| no | VLDL_P | 0 | 0 t-test | 1.016 | 0.022 | 0.111 | 0.005 |
| no | VLDL_PL | 0.461 | 0.467 t-test | 1.013 | 0.019 | 0.07 | 0.005 |
| no | VLDL_size | 38.998 | 39.008 t-test | 1 | 0 | 0.014 | 0.002 |
| no | VLDL_TG | 0.973 | 0.967 t-test | 0.994 | -0.009 | 0.018 | 0.002 |
| no | XL_HDL_C | 0.059 | 0.057 t-test | 0.968 | -0.047 | 0.31 | 0.06 |
| no | XL_HDL_CE | 0.042 | 0.04 t-test | 0.956 | -0.066 | 0.391 | 0.06 |
| no | XL_HDL_CE_pct | 40.214 | 33.187 t-test | 0.825 | -0.277 | 0.605 | 0.06 |
| no | XL_HDL_C_pct | 58.772 | 46.379 t-test | 0.789 | -0.342 | 0.52 | 0.06 |
| no | XL_HDL_FC | 0.016 | 0.016 t-test | 1.001 | 0.002 | 0.009 | 0.002 |
| no | XL_HDL_FC_pct | 18.557 | 13.192 t-test | 0.711 | -0.492 | 0.429 | 0.06 |
| no | XL_HDL_L | 0.105 | 0.106 t-test | 1.008 | 0.011 | 0.052 | 0.005 |
| no | XL_HDL_P | 0 | 0 t-test | 0.985 | -0.022 | 0.141 | 0.01 |
| no | XL_HDL_PL | 0.041 | 0.043 t-test | 1.053 | 0.074 | 0.239 | 0.06 |
| no | XL_HDL_PL_pct | 33.404 | 33.946 t-test | 1.016 | 0.023 | 0.143 | 0.01 |
| no | XL_HDL_TG | 0.006 | 0.006 t-test | 1.095 | 0.131 | 0.319 | 0.06 |
| no | XL_HDL_TG_pct | 7.824 | 5.389 t-test | 0.689 | -0.538 | 0.301 | 0.06 |
| no | XL_VLDL_C | 0.054 | 0.055 t-test | 1.019 | 0.027 | 0.072 | 0.005 |
| no | XL_VLDL_CE | 0.033 | 0.033 t-test | 1.024 | 0.034 | 0.119 | 0.005 |
| no | XL_VLDL_CE_pct | 18.462 | 17.45 t-test | 0.945 | -0.081 | 0.188 | 0.031 |
| no | XL_VLDL_C_pct | 28.74 | 27.987 t-test | 0.974 | -0.038 | 0.109 | 0.005 |
| no | XL_VLDL_FC | 0.022 | 0.022 t-test | 1.012 | 0.017 | 0.03 | 0.002 |
| no | XL_VLDL_FC_pct | 10.278 | 10.537 t-test | 1.025 | 0.036 | 0.153 | 0.013 |
| no | XL_VLDL_L | 0.203 | 0.207 t-test | 1.024 | 0.034 | 0.062 | 0.005 |
| no | XL_VLDL_P | 0 | 0 t-test | 1.03 | 0.043 | 0.083 | 0.005 |
| no | XL_VLDL_PL | 0.036 | 0.036 t-test | 1.014 | 0.019 | 0.032 | 0.002 |
| no | XL_VLDL_PL_pct | 16.268 | 17.052 t-test | 1.048 | 0.068 | 0.342 | 0.06 |
| no | XL_VLDL_TG | 0.113 | 0.116 t-test | 1.03 | 0.042 | 0.065 | 0.005 |
| no | XL_VLDL_TG_pct | 54.992 | 54.962 t-test | 0.999 | -0.001 | 0.003 | 0.002 |
| no | XS VLDL C | 0.142 | 0.144 t-test | 1.018 | 0.026 | 0.137 | 0.01 |
| no | XS VLDL CE | 0.096 | 0.095 t-test | 0.992 | -0.011 | 0.053 | 0.005 |
| no | XS VLDL CE pct | 32.455 | 30.476 t-test | 0.939 | -0.091 | 1 | 0.00 |
| no | XS_VLDL_C_pct | 47.868 | 46.003 t-test | 0.961 | -0.057 | 0.812 | 0.06 |
| no | XS_VLDL_C_pct XS_VLDL_FC | 0.046 | 0.049 t-test | 1.073 | 0.102 | 0.693 | 0.06 |
| | XS_VLDL_FC XS_VLDL_FC | 15.413 | 15.527 t-test | 1.073 | 0.102 | 0.23 | 0.06 |
| no<br>no | XS_VLDL_FC_pct XS_VLDL_L | 0.293 | 0.313 t-test | 1.068 | 0.011 | 0.627 | 0.06 |
| | AN VIIII I | | | | | | 0.00 |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 24/28 |

| no | XS_VLDL_PL | 0.084 | 0.093 t-test | 1.104 | 0.143 | 0.918 | 0.06 |
|---|---|---|---|---|---|---|---|
| no | XS_VLDL_PL_pct | 28.565 | 29.508 t-test | 1.033 | 0.047 | 1.022 | 0.06 |
| no | XS_VLDL_TG | 0.067 | 0.076 t-test | 1.127 | 0.173 | 0.818 | 0.06 |
| no | XS_VLDL_TG_pct | 23.567 | 24.49 t-test | 1.039 | 0.055 | 0.322 | 0.06 |
| no | XXL_VLDL_C | 0.046 | 0.049 t-test | 1.084 | 0.116 | 0.161 | 0.018 |
| no | XXL_VLDL_CE | 0.028 | 0.032 t-test | 1.137 | 0.185 | 0.331 | 0.06 |
| no | XXL_VLDL_CE_pct | 23.207 | 26.711 t-test | 1.151 | 0.203 | 0.268 | 0.06 |
| no | XXL_VLDL_C_pct | 36.128 | 39.55 t-test | 1.095 | 0.131 | 0.171 | 0.026 |
| no | XXL_VLDL_FC | 0.018 | 0.018 t-test | 1.001 | 0.001 | 0.001 | 0.001 |
| no | XXL_VLDL_FC_pct | 12.921 | 12.839 t-test | 0.994 | -0.009 | 0.011 | 0.002 |
| no | XXL_VLDL_L | 0.156 | 0.149 t-test | 0.957 | -0.064 | 0.054 | 0.005 |
| no | XXL_VLDL_P | 0 | 0 t-test | 0.992 | -0.012 | 0.01 | 0.002 |
| no | XXL_VLDL_PL | 0.026 | 0.026 t-test | 0.986 | -0.021 | 0.017 | 0.002 |
| no | XXL_VLDL_PL_pct | 14.889 | 16.636 t-test | 1.117 | 0.16 | 0.527 | 0.06 |
| no | XXL_VLDL_TG | 0.084 | 0.074 t-test | 0.879 | -0.187 | 0.136 | 0.01 |
| no | XXL_VLDL_TG_pct | 34.697 | 43.814 t-test | 1.263 | 0.337 | 0.413 | 0.06 |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 25/28 |

Table 5: Comparative Analysis of Metabolomic Pre-test and Post-test Results for Probiotics Group Blood Samples

| | I | | al expression and | | | 4 | | |
|---|---|---|---|---|---|---|---|---|
| Significance(p-value) | Feature | Mean(after) | Mean(before) | | | Log2(FC) | -Log10(p-value) | -Log10(padj) |
| yes | Acetate | 0.017 | | | 1.156 | | | |
| yes | Gly | 0.263 | | | 1.123 | 0.167 | 1.447 | 0.407 |
| yes | HDL_size | 9.573 | 9.508 1 | t-test | 0.993 | -0.01 | | |
| yes | Lactate | 4.175 | 5.984 1 | t-test | 1.433 | 0.519 | 1.441 | 0.407 |
| yes | L_VLDL_CE_pct | 14.036 | 15.354 1 | t-test | 1.094 | 0.129 | 1.363 | 0.407 |
| yes | L_VLDL_C_pct | 28.119 | 29.999 1 | t-test | 1.067 | 0.093 | 1.505 | 0.407 |
| yes | L_VLDL_FC_pct | 14.083 | 14.645 | t-test | 1.04 | 0.056 | 1.643 | 0.421 |
| yes | L_VLDL_L | 0.563 | 0.48 1 | t-test | 0.853 | -0.229 | 1.334 | 0.407 |
| yes | L_VLDL_TG | 0.288 | 0.233 1 | t-test | 0.81 | -0.304 | 2.037 | 0.533 |
| yes | L_VLDL_TG_pct | 51.128 | 49.056 1 | t-test | 0.959 | -0.06 | 1.429 | 0.407 |
| yes | M_HDL_CE_pct | 37.7 | 39.269 1 | t-test | 1.042 | 0.059 | 2.902 | 0.805 |
| yes | M HDL C pct | 46.11 | | | 1.03 | 0.043 | | 0.805 |
| yes | M_HDL_PL_pct | 47.018 | | | 0.986 | | | |
| yes | M HDL TG pct | 6.873 | | | 0.894 | -0.161 | | |
| yes | M_VLDL_PL_pct | 21.414 | | | 1.029 | 0.042 | | |
| yes | S HDL CE pct | 27.533 | | | 1.05 | 0.07 | | |
| yes | S_HDL_C_pct | 37.973 | | | 1.036 | | | |
| yes | S_HDL_PL_pct | 55.964 | | | 0.983 | -0.024 | | |
| | | 6.063 | | | 0.928 | -0.024 | | 0.407 |
| yes | S_HDL_TG_pct | 62.862 | | | | 0.019 | | |
| yes | S_LDL_C_pct | | | | 1.014 | | | |
| yes | TG_by_PG | 0.778 | | | 0.895 | -0.161 | | |
| yes | VLDL_size | 39.666 | | | 0.988 | | | |
| yes | VLDL_TG | 1.623 | | | 0.853 | -0.229 | | |
| yes | XL_HDL_CE_pct | 36.249 | | | 1.061 | 0.085 | | |
| yes | XL_HDL_C_pct | 52.182 | | | 1.081 | 0.113 | | |
| yes | XL_VLDL_L | 0.381 | | | 0.847 | -0.239 | | |
| yes | XL_VLDL_TG | 0.221 | | | 0.818 | | | |
| yes | XXL_VLDL_L | 0.467 | 0.375 1 | t-test | 0.804 | -0.315 | | 0.407 |
| yes | XXL_VLDL_P | 0 | 0 1 | t-test | 0.817 | -0.292 | | |
| yes | XXL_VLDL_TG | 0.267 | 0.202 1 | t-test | 0.756 | -0.403 | 2.073 | 0.533 |
| no | Acetoacetate | 0.026 | 0.017 | t-test | 0.651 | -0.619 | 0.697 | 0.243 |
| no | Acetone | 0.016 | 0.02 1 | t-test | 1.238 | 0.308 | 0.6 | 0.219 |
| no | Ala | 0.373 | 0.401 | t-test | 1.074 | 0.103 | 0.738 | 0.264 |
| no | Albumin | 41.766 | 43.735 1 | t-test | 1.047 | 0.066 | 1.025 | 0.384 |
| no | ApoA1 | 1.521 | 1.487 | t-test | 0.978 | -0.032 | 0.18 | 0.068 |
| no | АроВ | 1.001 | 1.016 | t-test | 1.015 | 0.021 | 0.123 | 0.039 |
| no | ApoB_by_ApoA1 | 0.669 | 0.698 1 | t-test | 1.044 | 0.062 | 0.667 | 0.227 |
| no | bOHbutyrate | 0.074 | 0.09 t | t-test | 1.218 | 0.284 | 0.375 | 0.158 |
| no | Cholines | 2.989 | | | 0.963 | -0.054 | | |
| no | Citrate | 0.062 | | | 1.012 | 0.017 | | |
| no | Clinical_LDL_C | 2.854 | | t-test | 1.051 | 0.072 | | |
| no | Creatinine | 72.354 | | | 0.949 | -0.075 | | |
| no | DHA | 0.287 | | | 0.94 | -0.09 | | |
| no | DHA_pct | 1.763 | | | 1.056 | 0.079 | | |
| | Gln | 0.546 | | | 1.006 | | | |
| no | | 4.989 | | | | | | |
| no | Glucose | | | | 0.89 | | | |
| no | GlycA | 0.94 | | | 0.998 | | | |
| no | Glycerol | 0.099 | | | 1.202 | | | |
| no | HDL_C | 1.29 | | | 0.978 | | | |
| no | HDL_CE | 0.986 | | | 0.985 | | | |
| no | HDL_FC | 0.303 | | | 0.957 | -0.063 | | |
| no | HDL_L | 3.102 | | | 0.962 | -0.056 | | |
| no | HDL_P | 0.016 | | t-test | 0.997 | | | |
| no | HDL_PL | 1.592 | 1.515 1 | t-test | 0.952 | -0.071 | 0.39 | 0.158 |
| no | HDL_TG | 0.22 | 0.208 1 | t-test | 0.942 | -0.085 | 0.361 | 0.158 |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 26/28 |

| no | His | 0.075 | 0.083 | t-test | 1.115 | 0.157 | 0.962 | 0.364 |
|---|---|---|---|---|---|---|---|---|
| no | IDL C | 0.867 | | t-test | 0.997 | -0.004 | 0.022 | 0.004 |
| no | IDL CE | 0.654 | | t-test | 0.991 | -0.013 | 0.086 | 0.027 |
| no | IDL CE pct | 49.557 | 49.108 | | 0.991 | -0.013 | 0.588 | 0.219 |
| no | IDL C pct | 65.567 | 65.379 | | 0.997 | -0.004 | 0.198 | 0.074 |
| no | IDL FC | 0.212 | | t-test | 1.018 | 0.025 | 0.156 | 0.057 |
| no | IDL FC pct | 16.01 | 16.271 | | 1.016 | 0.023 | 0.405 | 0.158 |
| no | IDL_L | 1.321 | | t-test | 1.004 | 0.006 | 0.036 | 0.004 |
| no | IDL P | 0 | | t-test | 0.96 | -0.059 | 0.352 | 0.158 |
| no | IDL PL | 0.305 | | t-test | 1.026 | 0.036 | 0.298 | 0.127 |
| no | IDL PL pct | 23.096 | 23.591 | | 1.021 | 0.031 | 0.914 | 0.337 |
| no | IDL_TG | 0.149 | | t-test | 0.998 | -0.003 | 0.013 | 0.004 |
| no | IDL TG pct | 11.338 | | t-test | 0.973 | -0.04 | 0.297 | 0.127 |
| no | lle | 0.072 | | t-test | 1.053 | 0.074 | 0.458 | 0.179 |
| no | LA | 5.312 | | t-test | 0.944 | -0.083 | 0.6 | 0.219 |
| no | LA_pct | 33.147 | 34.014 | | 1.026 | 0.037 | 0.435 | 0.172 |
| no | LDL C | 2.043 | | t-test | 1.025 | 0.064 | 0.627 | 0.172 |
| no | LDL CE | 1.542 | | t-test | 1.039 | 0.055 | 0.518 | 0.189 |
| no | LDL FC | 0.5 | | t-test | 1.064 | 0.033 | 0.967 | 0.169 |
| no | LDL L | 2.992 | | t-test | 1.004 | 0.056 | 0.496 | 0.304 |
| no | LDL P | 0.001 | | t-test | 1.035 | 0.05 | 0.367 | 0.154 |
| no | LDL_P | 0.714 | | t-test | 1.035 | 0.052 | 0.43 | 0.138 |
| no | LDL_PL | 23.826 | 23.839 | | 1.001 | 0.052 | 0.43 | 0.172 |
| no | LDL_Size | 0.235 | | t-test | 1.001 | 0.001 | 0.013 | 0.073 |
| | Leu | 0.142 | | t-test | 1.101 | 0.003 | 1.113 | 0.396 |
| no | L HDL C | 0.142 | | t-test | 0.881 | -0.183 | 0.507 | 0.396 |
| no | L HDL CE | 0.239 | | t-test | 0.889 | -0.169 | 0.455 | 0.189 |
| no | L HDL CE pct | 30.952 | | t-test | 1.059 | 0.083 | 0.455 | 0.179 |
| | L_HDL_C_pct | 40.163 | 41.444 | | 1.039 | 0.085 | 0.471 | 0.183 |
| no | L HDL FC | 0.057 | | t-test | 0.855 | -0.226 | 0.471 | 0.163 |
| no | | 9.212 | | t-test | 0.833 | -0.226 | 1.2 | 0.242 |
| no | L_HDL_FC_pct<br>L HDL L | 0.575 | | t-test | 0.939 | -0.184 | 0.564 | 0.407 |
| | | 0.001 | | | | -0.184 | 0.504 | |
| no | L_HDL_P | | | t-test | 0.876 | | | 0.189 |
| no | L_HDL_PL | 0.289<br>51.142 | | t-test | 0.873 | -0.196<br>-0.035 | 0.643<br>1.046 | 0.224<br>0.384 |
| no | L_HDL_PL_pct | | 49.923 | | 0.976 | | | |
| no | L_HDL_TG | 0.046 | | t-test | 0.921 | -0.119 | 0.359 | 0.158 |
| no | L_HDL_TG_pct | 8.695 | | t-test | 0.993 | -0.01 | 0.027 | 0.004 |
| no | L_LDL_C | 1.274 | | t-test | 1.046 | 0.064 | 0.644 | 0.224 |
| no | L_LDL_CE | 0.961 | | t-test | 1.042 | 0.059 | 0.575 | 0.219 |
| no | L_LDL_CE_pct | 52.644 | 52.638 | | 1 | 0 | 0.007 | 0.004 |
| no | L_LDL_C_pct | 69.77 | 70.032 | | 1.004 | 0.005 | 0.282 | 0.122 |
| no | L_LDL_FC | 0.313 | | t-test | 1.057 | 0.08 | 0.859 | 0.308 |
| no | L_LDL_FC_pct | 17.127 | 17.394 | | 1.016 | 0.022 | 0.781 | 0.275 |
| no | L_LDL_L | 1.825 | | t-test | 1.043 | 0.06 | 0.556 | 0.214 |
| no | L_LDL_P | 0.001 | | t-test | 1.042 | 0.06 | 0.401 | 0.158 |
| no | L_LDL_PL | 0.4 | | t-test | 1.044 | 0.062 | 0.555 | 0.214 |
| no | L_LDL_PL_pct | 21.932 | | t-test | 1.001 | 0.001 | 0.054 | 0.013 |
| no | L_LDL_TG | 0.151 | | t-test | 1.015 | 0.021 | 0.089 | 0.027 |
| no | L_LDL_TG_pct | 8.298 | | t-test | 0.966 | -0.05 | 0.355 | 0.158 |
| no | L_VLDL_C | 0.155 | | t-test | 0.912 | -0.132 | 0.51 | 0.189 |
| no | L_VLDL_CE | 0.075 | | t-test | 0.932 | -0.102 | 0.326 | 0.144 |
| no | L_VLDL_FC | 0.08 | | t-test | 0.894 | -0.162 | 0.742 | 0.264 |
| no | L_VLDL_P | 0 | | t-test | 0.866 | -0.208 | 1.116 | 0.396 |
| no | L_VLDL_PL | 0.12 | | t-test | 0.879 | -0.186 | 0.933 | 0.348 |
| no | L_VLDL_PL_pct | 20.753 | | t-test | 1.009 | 0.013 | 0.269 | 0.114 |
| no | M_HDL_C | 0.496 | | t-test | 0.984 | -0.023 | 0.094 | 0.027 |
| no | M_HDL_CE | 0.404 | | t-test | 0.991 | -0.013 | 0.053 | 0.013 |
| no | M_HDL_FC | 0.092 | | t-test | 0.954 | -0.068 | 0.272 | 0.115 |
| no | M_HDL_FC_pct | 8.409 | | t-test | 0.981 | -0.028 | 0.83 | 0.307 |
| no | M_HDL_L | 1.091 | | t-test | 0.968 | -0.048 | 0.219 | 0.086 |
| no | M_HDL_P | 0.004 | 0.004 | t-test | 0.967 | -0.048 | 0.201 | 0.074 |
| no | M_HDL_PL | 0.515 | 0.493 | t-test | 0.957 | -0.063 | 0.329 | 0.144 |
| no | M_HDL_TG | 0.08 | 0.074 | t-test | 0.931 | -0.102 | 0.427 | 0.172 |
| no | M_LDL_C | 0.544 | 0.57 | t-test | 1.048 | 0.068 | 0.625 | 0.222 |
| no | M_LDL_CE | 0.408 | 0.424 | t-test | 1.038 | 0.054 | 0.47 | 0.183 |
| no | M_LDL_CE_pct | 50.244 | EO 190 | t-test | 0.999 | -0.002 | 0.047 | 0.009 |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 27/28 |

| | leaves a constitution | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| no | M_LDL_C_pct | 67.302 | 67.855 | | 1.008 | 0.012 | 0.601 | 0.219 |
| no | M_LDL_FC | 0.136 | | t-test | 1.079 | 0.109<br>0.051 | 1.039 | 0.384 |
| no | M_LDL_FC_pct | 17.057<br>0.809 | 17.667 | t-test | 1.036 | 0.051 | 1.151<br>0.474 | 0.407<br>0.183 |
| no | M_LDL_L<br>M_LDL_P | 0.809 | | | 1.042<br>1.028 | 0.039 | 0.474 | 0.183 |
| no | M LDL PL | 0.209 | | t-test<br>t-test | 1.028 | 0.059 | 0.365 | 0.123 |
| no<br>no | M LDL PL pct | 25.892 | 25.737 | | 0.994 | -0.009 | 0.322 | 0.138 |
| no | M LDL TG | 0.057 | | t-test | 0.995 | -0.003 | 0.025 | 0.144 |
| | M LDL TG pct | 6.806 | | t-test | 0.995 | -0.007 | 0.703 | 0.004 |
| no<br>no | MUFA | 4.058 | | t-test | 0.941 | -0.087 | 0.703 | 0.245 |
| no | MUFA_pct | 24.27 | 23.809 | | 0.94 | -0.089 | 0.376 | 0.219 |
| no | M VLDL C | 0.186 | | t-test | 1.032 | 0.046 | 0.145 | 0.158 |
| no | M VLDL CE | 0.088 | | t-test | 1.091 | 0.126 | 0.459 | 0.032 |
| no | M VLDL CE pct | 12.017 | 14.183 | | 1.18 | 0.120 | 1.276 | 0.407 |
| no | M_VLDL_C_pct | 24.376 | 27.164 | | 1.114 | 0.156 | 1.262 | 0.407 |
| no | M VLDL FC | 0.098 | | t-test | 0.979 | -0.03 | 0.092 | 0.407 |
| no | M VLDL FC pct | 12.359 | 12.981 | | 1.05 | 0.071 | 1.168 | 0.407 |
| no | M VLDL L | 0.816 | | t-test | 0.934 | -0.099 | 0.434 | 0.407 |
| no | M VLDL P | 0.810 | | t-test | 0.954 | -0.068 | 0.265 | 0.112 |
| no | M VLDL PL | 0.172 | | t-test | 0.963 | -0.055 | 0.195 | 0.112 |
| no | M_VLDL_TG | 0.457 | | t-test | 0.883 | -0.033 | 0.193 | 0.364 |
| no | M_VLDL_TG_pct | 54.21 | 50.792 | | 0.883 | -0.18 | 1.284 | 0.304 |
| no | non_HDL_C | 3.838 | | t-test | 1.018 | 0.026 | 0.159 | 0.407 |
| no | Omega_3 | 0.782 | | t-test | 0.881 | -0.183 | 0.48 | 0.037 |
| no | Omega_3_pct | 4.53 | | t-test | 0.881 | -0.183 | 0.325 | 0.144 |
| no | Omega 6 | 6.048 | | t-test | 0.953 | -0.069 | 0.581 | 0.144 |
| no | Omega_6_by_Omega_3 | 9.266 | 10.779 | | 1.163 | 0.218 | 0.864 | 0.308 |
| no | Omega 6 pct | 38.082 | 39.375 | | 1.034 | 0.048 | 0.837 | 0.308 |
| no | Phe | 0.085 | | t-test | 1.011 | 0.048 | 0.12 | 0.038 |
| no | Phosphatidylc | 2.461 | | t-test | 0.944 | -0.084 | 0.612 | 0.038 |
| no | Phosphoglyc | 2.716 | | t-test | 0.955 | -0.066 | 0.441 | 0.213 |
| no | PUFA | 6.83 | | t-test | 0.935 | -0.081 | 0.636 | 0.173 |
| no | PUFA by MUFA | 1.789 | | t-test | 1.049 | 0.069 | 0.571 | 0.218 |
| no | PUFA pct | 42.612 | 43.651 | | 1.024 | 0.035 | 0.58 | 0.218 |
| no | Pyruvate | 0.04 | | t-test | 1.456 | 0.542 | 0.37 | 0.158 |
| no | Remnant C | 1.796 | | t-test | 0.988 | -0.018 | 0.079 | 0.026 |
| no | SFA | 5.491 | | t-test | 0.941 | -0.088 | 0.472 | 0.183 |
| no | SFA_pct | 33.118 | | t-test | 0.983 | -0.025 | 0.505 | 0.189 |
| no | S HDL C | 0.486 | | t-test | 1.029 | 0.041 | 0.354 | 0.158 |
| no | S_HDL_CE | 0.351 | | t-test | 1.038 | 0.054 | 0.534 | 0.130 |
| no | S HDL FC | 0.135 | | t-test | 1.005 | 0.007 | 0.042 | 0.008 |
| no | S_HDL_FC_pct | 10.441 | 10.436 | | 1 | -0.001 | 0.017 | 0.004 |
| no | S HDL L | 1.295 | | t-test | 1.004 | 0.005 | 0.03 | 0.004 |
| no | S HDL P | 0.011 | | t-test | 1.025 | 0.035 | 0.284 | 0.122 |
| no | S HDL PL | 0.727 | | t-test | 0.991 | -0.013 | 0.079 | 0.026 |
| no | S HDL TG | 0.082 | | t-test | 0.967 | -0.049 | 0.238 | 0.1 |
| no | S_LDL_C | 0.225 | | t-test | 1.035 | 0.05 | 0.388 | 0.158 |
| no | S LDL CE | 0.173 | | t-test | 1.026 | 0.037 | 0.24 | 0.1 |
| no | S LDL CE pct | 48.121 | | t-test | 1.004 | 0.005 | 0.188 | 0.073 |
| no | S LDL FC | 0.051 | | t-test | 1.067 | 0.093 | 1.031 | 0.384 |
| no | S LDL FC pct | 14.741 | 15.416 | | 1.046 | 0.065 | 0.854 | 0.304 |
| no | S LDL L | 0.358 | | t-test | 1.021 | 0.029 | 0.212 | 0.081 |
| no | S LDL P | 0.558 | | t-test | 1.021 | 0.023 | 0.194 | 0.074 |
| no | S LDL PL | 0.106 | | t-test | 1.009 | 0.012 | 0.089 | 0.027 |
| no | S_LDL_PL_pct | 29.648 | | t-test | 0.991 | -0.013 | 0.371 | 0.158 |
| no | S LDL TG | 0.028 | | t-test | 0.948 | -0.076 | 0.358 | 0.158 |
| no | S LDL TG pct | 7.49 | | t-test | 0.922 | -0.070 | 0.774 | 0.138 |
| no | Sphingomyelins | 0.477 | | t-test | 0.989 | -0.117 | 0.088 | 0.027 |
| no | S_VLDL_C | 0.199 | | t-test | 1.033 | 0.047 | 0.162 | 0.027 |
| no | S_VLDL_CE | 0.126 | | t-test | 1.033 | 0.047 | 0.102 | 0.037 |
| no | S_VLDL_CE<br>S_VLDL_CE_pct | 21.368 | 22.914 | | 1.072 | 0.101 | 1.147 | 0.407 |
| no | S_VLDL_C_pct | 33.978 | | t-test | 1.072 | 0.101 | 1.147 | 0.407 |
| no | S_VLDL_C_pct<br>S_VLDL_FC | 0.073 | | t-test | 1.022 | 0.031 | 0.105 | 0.407 |
| | J VLDL I C | 0.073 | | | 1.044 | 0.031 | 0.103 | 0.03 |
| no | S_VLDL_FC_pct | 12.61 | | t-test | 1.07 | 0.097 | 1.238 | 0.407 |

| IRB/REC No.: | CMUH110-REC2<br>-070 |
|--------------|----------------------|
| Page No.: | 28/28 |

| no | S_VLDL_P | 0 | 0 | t-test | 0.966 | -0.05 | 0.165 | 0.057 |
|---|---|---|---|---|---|---|---|---|
| no | S VLDL PL | 0.133 | | t-test | 0.998 | -0.003 | 0.008 | 0.004 |
| no | S_VLDL_PL_pct | 22.398 | 23.208 | | 1.036 | 0.051 | 1.163 | 0.407 |
| no | S VLDL TG | 0.279 | | t-test | 0.922 | -0.117 | 0.453 | 0.179 |
| no | S VLDL TG pct | 43.624 | 40.388 | | 0.926 | -0.111 | 1.19 | 0.407 |
| no | Total_BCAA | 0.486 | | t-test | 1.071 | 0.099 | 0.842 | 0.308 |
| no | Total_C | 5.128 | 5.17 | t-test | 1.008 | 0.012 | 0.07 | 0.024 |
| no | Total_CE | 3.693 | 3.734 | t-test | 1.011 | 0.016 | 0.1 | 0.028 |
| no | Total_FA | 16.38 | 15.438 | t-test | 0.943 | -0.085 | 0.618 | 0.22 |
| no | Total_FC | 1.435 | 1.436 | t-test | 1.001 | 0.001 | 0.005 | 0.003 |
| no | Total_L | 10.668 | 10.37 | t-test | 0.972 | -0.041 | 0.248 | 0.103 |
| no | Total_P | 0.018 | 0.018 | t-test | 0.999 | -0.001 | 0.008 | 0.004 |
| no | Total_PL | 3.313 | 3.224 | t-test | 0.973 | -0.039 | 0.239 | 0.1 |
| no | Total_TG | 2.227 | 1.976 | t-test | 0.887 | -0.172 | 1.011 | 0.384 |
| no | Tyr | 0.066 | 0.07 | t-test | 1.046 | 0.065 | 0.448 | 0.177 |
| no | Unsaturation | 1.369 | 1.37 | t-test | 1 | 0.001 | 0.018 | 0.004 |
| no | Val | 0.272 | 0.288 | t-test | 1.06 | 0.084 | 0.657 | 0.227 |
| no | VLDL_C | 0.929 | 0.909 | t-test | 0.978 | -0.031 | 0.107 | 0.03 |
| no | VLDL_CE | 0.523 | 0.526 | t-test | 1.004 | 0.006 | 0.02 | 0.004 |
| no | VLDL_FC | 0.406 | 0.383 | t-test | 0.945 | -0.082 | 0.314 | 0.139 |
| no | VLDL_L | 3.254 | 2.949 | t-test | 0.906 | -0.142 | 0.708 | 0.245 |
| no | VLDL_P | 0 | 0 | t-test | 0.958 | -0.063 | 0.261 | 0.111 |
| no | VLDL_PL | 0.702 | 0.655 | t-test | 0.934 | -0.099 | 0.411 | 0.159 |
| no | XL_HDL_C | 0.068 | 0.062 | t-test | 0.918 | -0.123 | 0.731 | 0.262 |
| no | XL_HDL_CE | 0.049 | 0.044 | t-test | 0.909 | -0.138 | 0.636 | 0.224 |
| no | XL_HDL_FC | 0.019 | 0.018 | t-test | 0.943 | -0.085 | 0.756 | 0.264 |
| no | XL_HDL_FC_pct | 15.933 | 17.975 | t-test | 1.128 | 0.174 | 0.844 | 0.308 |
| no | XL_HDL_L | 0.141 | 0.123 | t-test | 0.875 | -0.193 | 0.897 | 0.331 |
| no | XL_HDL_P | 0 | 0 | t-test | 0.913 | -0.132 | 0.662 | 0.227 |
| no | XL_HDL_PL | 0.06 | 0.049 | t-test | 0.814 | -0.297 | 1.022 | 0.384 |
| no | XL_HDL_PL_pct | 37.258 | 33.048 | t-test | 0.887 | -0.173 | 1.267 | 0.407 |
| no | XL_HDL_TG | 0.012 | 0.012 | t-test | 0.933 | -0.1 | 0.376 | 0.158 |
| no | XL_HDL_TG_pct | 10.56 | 10.531 | | 0.997 | -0.004 | 0.015 | 0.004 |
| no | XL_VLDL_C | 0.089 | | t-test | 0.918 | -0.124 | 0.471 | 0.183 |
| no | XL_VLDL_CE | 0.047 | | t-test | 0.966 | -0.05 | 0.149 | 0.054 |
| no | XL_VLDL_CE_pct | 14.714 | 17.751 | | 1.206 | 0.271 | 1.142 | 0.407 |
| no | XL_VLDL_C_pct | 25.817 | 29.087 | | 1.127 | 0.172 | 1.084 | 0.385 |
| no | XL_VLDL_FC | 0.041 | | t-test | 0.863 | -0.213 | 0.988 | 0.368 |
| no | XL_VLDL_FC_pct | 11.103 | 11.336 | | 1.021 | 0.03 | 0.48 | 0.183 |
| no | XL_VLDL_P | 0 | | t-test | 0.857 | -0.222 | 1.223 | 0.407 |
| no | XL_VLDL_PL | 0.071 | | t-test | 0.851 | -0.232 | 1.151 | 0.407 |
| no | XL_VLDL_PL_pct | 18.5 | 18.311 | | 0.99 | -0.015 | 0.376 | 0.158 |
| no | XL_VLDL_TG_pct | 55.683 | 52.602 | | 0.945 | -0.082 | 1.051 | 0.384 |
| no | XS_VLDL_C | 0.183 | | t-test | 1.01 | 0.014 | 0.074 | 0.024 |
| no | XS_VLDL_CE | 0.12 | | t-test | 1.015 | 0.021 | 0.137 | 0.049 |
| no | XS_VLDL_CE_pct | 29.837 | 31.525 | | 1.057 | 0.079 | 1.028 | 0.384 |
| no | XS_VLDL_C_pct | 44.926 | 46.821 | | 1.042 | 0.06 | 1.089 | 0.385 |
| no | XS_VLDL_FC | 0.062 | | t-test | 1 014 | 0.001 | 0.003 | 0.003 |
| no | XS_VLDL_FC_pct | 15.089 | 15.296 | | 1.014 | 0.02<br>-0.011 | 0.738<br>0.045 | 0.264 |
| no | XS_VLDL_L | 0.417 | | t-test | 0.992 | -0.011 | 0.045 | 0.009<br>0.004 |
| no | XS_VLDL_P | | | t-test | 0.997 | -0.005 | 0.021 | |
| no | XS_VLDL_PL | 0.124<br>29.481 | 28.941 | t-test | 0.985 | -0.021 | | 0.026<br>0.264 |
| no | XS_VLDL_PL_pct | 0.111 | | | 0.982<br>0.971 | -0.027 | 0.738<br>0.157 | |
| no | XS_VLDL_TG XS_VLDL_TG pct | 25.593 | | t-test<br>t-test | 0.947 | -0.042 | 0.157 | 0.057<br>0.337 |
| no | XXL VLDL_IG_pct | 0.118 | | t-test | 0.947 | -0.078 | 0.589 | 0.337 |
| no<br>no | XXL_VLDL_CE | 0.118 | | t-test | 0.885 | -0.177 | 0.372 | 0.219 |
| no | XXL_VLDL_CE_pct | 17.383 | | t-test | 1.084 | 0.116 | 0.223 | 0.138 |
| no | XXL_VLDL_C_pct | 28.919 | 30.122 | | 1.042 | 0.110 | 0.106 | 0.088 |
| no | XXL_VLDL_C_ptt | 0.051 | | t-test | 0.847 | -0.239 | 0.100 | 0.348 |
| no | XXL_VLDL_FC_pct | 11.537 | 11.284 | | 0.847 | -0.239 | 0.055 | 0.013 |
| no | XXL_VLDL_PL | 0.082 | | t-test | 0.842 | -0.032 | 1.017 | 0.013 |
| no | XXL_VLDL_PL_pct | 17.037 | 16.536 | | 0.842 | -0.248 | 0.081 | 0.026 |
| no | XXL VLDL_FL_pct | 54.043 | 42.231 | | 0.781 | -0.043 | 1.188 | 0.020 |
| | ///r_v_bbt_10_pct | 34.043 | -12.231 | | 0.701 | 0.550 | 1.100 | 0.407 |